# **CLINICAL STUDY PROTOCOL**

Virologic Outcomes of Lamivudine/Dolutegravir in Virologically suppressed subjects with Expected or confirmed Resistance to Lamivudine (VOLVER Study)

Sponsor: Fundación SEIMC-GESIDA

Protocol code: GESIDA 11820

Nº EduraCT: 2021-000290-84

**Sponsor Contact:** C/ Agustín de Betancourt, 13-Entreplanta. 28003, Madrid (Spain)

Tel: +34 91 556 80 25

Version of Protocol: 4.0

Date of Protocol: 31. May. 2021



# **Confidential information**

This protocol contains confidential information; therefore, it should be considered as confidential and limited to its intended use in this clinical trial. This protocol is only to be disclosed to the staff of Fundación SEIMC-GESIDA; Health Authorities; staff in charge of the review, authorisation, monitoring, auditing or inspection of the clinical trial; and also to the clinical staff in charge of conducting it. This material is not to be disclosed to individuals outside of this clinical trial without prior written authorisation from Fundación SEIMC-GESIDA.



# PROTOCOL SIGNATURE PAGE

**Study Title:** Virologic Outcomes of Lamivudine/Dolutegravir in Virologically suppressed subjects with Expected or confirmed Resistance to Lamivudine (VOLVER study).

**Protocol Code:** GESIDA 11820 **EudraCT No.:** 2021-000290-84 **Version:** 4.0 of 31 May 2021

Sponsor: Fundación SEIMC - GESIDA

| Signature of the Coordinating Investigators: | | |
|---|---|---|
| Dr José Ramón Arribas - L | a Paz University Hospital | |
| Name | <br>Signature | <br>Date |
| | Ç | |
| Dr Federico Pulido - 12 de | Octubre Hospital | |
| Name | Signature | Date |
| Signature of the sponsor | | |
| Dr Juan Julián Gonzalez G | arcía - Chairperson of the Board | d of Directors |
| Name | Signature | Date |
| Signature of the Principa | Investigator: | |
| Name: | Site: | |
| Name | <br>Signature | |





#### 1. SUMMARY

I. Sponsor: Fundación SEIMC-GESIDA

**II. Clinical study title:** Virologic Outcomes of Lamivudine/Dolutegravir in Virologically suppressed subjects with Expected or confirmed Resistance to Lamivudine (VOLVER study).

### III. Principal Investigators:

Dr. José Ramón Arribas López

La Paz University Hospital.

Internal Medicine Department. Infectious Diseases Unit.

Paseo de la Castellana, 261. CP 28046 - Madrid

e-mail: joser.arribas@salud.madrid.org

Dr. Federico Pulido

12 de Octubre University Hospital.

Internal Medicine Department. HIV Unit.

Centro de Actividades Ambulatorias 2ª Planta Bloque D.

Av. Cordoba s/n. 28041-Madrid

e-mail: federico.pulido@salud.madrid.org

# IV. Clinical study phase: Ila.

# V. Team participants:

Multicentre study, to be conducted at 17 healthcare centres in Spain. The listing of all investigators and sites will be attached in a separate document.

#### VI. Background:

Dolutegravir (DTG) plus lamivudine (3TC) is a dual regimen combination recommended for both naïve and suppressed persons with HIV-1 infection<sup>1</sup>. However, data regarding the efficacy of this regimen in suppressed persons with history of past resistance or virologic failures is currently insufficient. In particular, it is important to determine if this combination is safe to use in persons with past resistance to 3TC. Limited data from retrospective cohorts, and a small number of participants from the DOLULAM and TANGO studies seem to point that DTG/3TC may be used without exposing individuals



to a significant risk of virologic failure, despite historical 3TC resistance or archived minority 3TC resistance-associated mutations <sup>2-5</sup>. In our prospective pilot study ART-PRO<sup>6</sup> 18/21 persons with past M184V/I mutations, not detected at baseline through proviral DNA Sanger sequencing, were switched to DTG/3TC and maintained virologic control for 96 weeks without any case of virologic failure<sup>7</sup>. In our study, archived 3TCresistance associated mutations were detected at baseline through next-generation sequencing (NGS) over the 5% threshold in more than half of participants with past 3TC resistance, without any detrimental effect on viral control. Although showing promising results, ART PRO study's generalizability is limited due to the small size and the exclusion of participants exposed to integrase inhibitors, which call for a larger study. VOLVER study aims to enrol persons with confirmed or suspected history of 3TC resistance and demonstrate that, when proviral DNA population sequencing no longer detects 3TC resistance-associated mutations, DTG/3TC is sufficient to maintain virologic suppression. Based in our prior findings, we also want to confirm that the virological impact of 3TC-resistant archived minority variants prior to switching to DTG/3TC is negligible in this context.

### VII. Study design:

Phase IIa, open-label, single arm, multicentric study. Follow up: 96 weeks.

#### VIII. Study treatment:

Dovato® (Dolutegravir 50 mg/Lamivudine 300 mg film-coated tablet):

Route of administration: oral.

Dose: Dolutegravir 50 mg/Lamivudine 300 mg/day.

Posology: one 50 mg/300 mg film coated-tablet once daily.

Intervention: change of current antiretroviral treatment to DTG 50 mg/3TC 300 mg QD.

#### IX. Study Locations:

This is a multicentre study, and it will be conducted at different healthcare centres in Spain. The listing of all investigators and sites where the clinical trial is going to be conducted is attached in a separate document

### X. Estimated sample size:



120 participants. A minimum of 30%-50% of the study population would be required to have historical RNA population genotype with confirmed M184V/I mutation.

#### XI. Ethics Committee:

The study will be evaluated by the Ethics Committee (Comité de Ética de la Investigación con medicamentos) of University Hospital La Paz which is authorized by the Ministry of Health and Consumer Affairs (https://www.aemps.gob.es/investigacionClinica/medicamentos/docs/listado -comites-investigacion-clinica.pdf) and by the health authorities of the Autonomous Community of Madrid (Spain).

# XII. Hypothesis:

Our hypothesis is that therapy with DTG/3TC would be able to maintain viral control in HIV infected participants with prior history of 3TC resistance but without evidence of M184V/I resistance mutation in proviral DNA population sequencing at baseline. We also hypothesize that archived minority 3TC resistance associated mutations detected by next-generation (NGS) sequencing prior to the switch would not have a significant impact on the efficacy of DTG/3TC.

# XIII. Study Objectives and Endpoints:

| Primary objective | Primary endpoint |
|---|---|
| To assess the efficacy of a switch to DTG/3TC | Proportion of virologic failure (VF) defined as |
| for maintenance of virologic suppression at 48 | HIV-1 RNA viral load (VL) ≥ 50 copies per mL |
| weeks in persons with past confirmed or | at 48 weeks (in the intention-to-treat-exposed |
| suspected 3TC resistance, when proviral DNA | population (ITT-e) using the US Food and |
| population sequencing does not detect 3TC | Drug Administration (FDA) snapshot |
| resistance-associated mutations at baseline. | algorithm). |
| Secondary objectives | Secondary endpoints |
| | - Proportion of VF (≥50 copies/mL) at week |
| | 96, ITT-e, FDA snapshot. |
| To evaluate ather estimations of virological | - Proportion of VF (≥50 copies/mL) at week |
| To evaluate other estimations of virological | 48 and 96, per protocol population (PP), |
| control at weeks 48 and 96. | FDA snapshot. |
| | - Proportion of VF (≥200 copies/mL) at |
| | week 48 and 96, ITT-e and PP population, |

VOLVER Study protocol 4.0, 31 May 2021





| | FDA snapshot. |
|---|---|
| | - Proportion of Confirmed Virologic |
| | Withdrawal ([CVW]: A VL≥ 50 copies/mL |
| | followed by a VL≥ 200 copies/mL in re- |
| | test) at weeks 48 and 96, ITT-e and PP |
| | population, FDA snapshot. |
| | - Proportion of Precautionary Virologic |
| | Withdrawal ([PVW]: three consecutive VL |
| | between 50- 200 copies/mL) at weeks 48 |
| | and 96, ITT-e and PP population, FDA |
| | snapshot. |
| | - Proportion of participants with VL<50 |
| | copies/mL week 48 and 96, ITT-e and per |
| | protocol population, FDA snapshot. |
| To compare visual registers in norman | - Incidence of VF with drug resistance |
| To assess viral resistance in persons | associated mutations. |
| experiencing VF. | - Describe number and type of resistance- |
| | associated mutations in VF |
| | - Analysis of factors associated to VF (i.e |
| | time to VF). |
| | - Proportion of VF in pre-specified |
| | subgroups: |
| To evaluate factors associated with VF. | - Confirmed historical M184V/I vs No |
| | resistance mutations |
| | - INSTI exposure vs No prior INSTI |
| | exposure |
| | - Time virologically suppressed |
| | - Time on 3TC/FTC |
| | - Proportion of participants with VF with |
| To assess the impact of baseline archived | baseline 3TC or INSTI resistance- |
| minority 3TC resistance-associated mutations | associated mutations detected at |
| in viral control (in cases of VF and transient | baseline by NGS with 1, 5, and 20% |
| viral rebounds [VL≥50copies/mL preceded | threshold. |
| and followed by VL<50 copies/mL]). | - Proportion of participants with transient |
| | viral rebounds with baseline 3TC or INSTI |
| | viral repoditios with pasellile 310 of INSTI |



| | resistance- associated mutations |
|---|---|
| | detected at baseline by NGS with 1, 5, |
| | and 20% threshold. |
| To evaluate the dynamics of archived minority | Type and frequency of resistance mutations |
| 3TC resistance-associated mutations after | (RT and integrase) in proviral DNA measured |
| switching to DTG/3TC at 96 weeks. | by NGS at baseline and week 96. |
| To evaluate the immune effects of switch to | Change from Baseline in CD4+ cell count and |
| | in CD4+/CD8+ cell counts ratio at weeks 48 |
| DTG/3TC | and 96 |
| | - Incidence and severity of AEs and |
| | laboratory abnormalities through week 48 |
| To evaluate the safety and tolerability of | and 96. |
| DTG/3TC in this study | - Proportion of subjects who discontinue |
| | treatment due to AEs through weeks 48 |
| | and 96. |

# XIV. Disease under study: HIV-1 infection.

# XV. Study population:

Persons receiving antiretroviral treatment, followed at study participating centres.

# Inclusion Criteria:

- a. Adults (≥ 18 years old) with HIV-1 infection able to understand and give informed written consent.
- b. Stable ART in the 12 weeks prior to screening visit.
  - Only switch for tolerability/convenience/access reasons to generic drugs or switch from ritonavir to cobicistat or TDF to TAF would be allowed in the 12-week window and as long as the components of the regimen are unchanged.
- c. Viral load <50 copies/mL at screening and in the year prior to study entry.
  - A blip (50-500 copies/mL) would be allowed within 48 weeks prior to inclusion in the study, if preceded and followed by an undetectable VL determination.
- d. CD4<sup>+</sup> count > 200 cells/µL at screening.



- e. History of 3TC resistance: either *confirmed historical 3TC resistance* (historical RNA Sanger or RNA NGS>20% threshold genotype with M184V/I mutation) OR *suspected historical 3TC resistance*.
  - Suspicion of past 3TC resistance is defined as any of the following:
    - i. Previous treatment with only 2 NRTIs (1 of them being emtricitabine or 3TC [XTC]).
    - ii. Two consecutive VL > 200 copies/mL while on treatment including XTC.
    - iii. One VL > 200 copies/mL while on treatment including XTC <u>PLUS</u> change of ART as consequence of that elevated VL.

#### **Exclusion Criteria:**

- Participants with M184V/I or K65R in screening visit proviral DNA Sanger genotype.
- b. Prior virologic failure (VF) under integrase inhibitor (INSTI)- based regimen.
   defined as two consecutive VL > 200 copies/mL while receiving INSTI regardless of genotypic test results
- c. INSTI resistance mutations in historical RNA genotype.
- d. Documented resistance to DRV defined as the presence of a combination of mutations scored with at least 15 points in the Stanford University HIV Drug Resistance Database.
- e. Positive Surface Hepatitis B Ag (HBAgS) OR negative HBAgS and negative hepatitis B surface antibody (anti-HBs) with positive anti-core antibody (anti-HBc) and positive HBV DNA.
- f. Pregnant, breastfeeding women, women with a positive pregnancy test at the time of screening, sexually active fertile women wishing to conceive or unwilling to commit to contraceptive methods (see Appendix 1 for the accepted list of the highly effective methods for avoiding pregnancy), for the duration of the study and until 4 weeks after the last dose of study medication. All women are considered fertile unless they have undergone a sterilizing surgery or are over the age of 50 with spontaneous amenorrhea for over 12 months prior to study entry.



- g. Patients with active opportunistic infections or cancer requiring intravenous treatment and/or chemotherapy at screening.
- h. Any comorbidities or treatment with experimental drugs that according to the investigator could bias study results or entail additional risks for the participant.
- i. Participants receiving other medications that according to study drug label are contraindicated.
- j. Severe hepatic impairment (Class C) as determined by Child-Pugh classification.
- k. Alanine aminotransferase (ALT) over 5 times the upper limit of normal (ULN) or ALT over 3xULN and bilirubin over 1.5xULN.
- Unstable liver disease (as defined by the presence of ascites, encephalopathy, coagulopathy, hypoalbuminemia, oesophageal or gastric varices, or persistent jaundice), cirrhosis, known biliary abnormalities (apart from hyperbilirubinemia or jaundice due to Gilbert's syndrome or asymptomatic gallstones);
- m. Creatinine clearance of <30 mL/min/1.73m<sup>2</sup> via CKD-EPI method.
- n. Any verified Grade 4 laboratory abnormality that to the investigators criteria would affect the safety of the participant if included in the study.
- o. History or presence of allergy to dolutegravir or lamivudine.

# XVI. Duration of the study:

- i. Duration of the participant selection period: 9 months.
- ii. Duration of the follow-up period: 96 weeks.
- iii. Data analysis and preparation of the final report: 6 months.



# 2. INDEX

| 1. | SUMM | ARY | 3 |
|---|---|---|---|
| 2. | INDEX | | .10 |
| 3. | GENE | RAL INFORMATION | .14 |
| | 3.1 | Study identification | .14 |
| | 3.2 | Type of clinical study | .14 |
| | 3.2 | Study drug description | .14 |
| | 3.3 | Principal investigators | .14 |
| | 3.4 | Collaborating centres | .14 |
| | 3.5 | Monitor identification | .15 |
| | 3.6 | Ethics committee of reference identification | .15 |
| | 3.7 | Expected duration | .15 |
| 4. | BACK | GROUND AND JUSTIFICATION | .15 |
| 5. | нүро | THESIS AND OBJECTIVES | .17 |
| | 5.1 Hy | pothesis | .17 |
| | 5.2 Ob | jectives | .18 |
| 6. | TYPE | OF CLINICAL STUDY AND DESIGN | .20 |
| | 6.1 Clii | nical study phase | .20 |
| | 6.2 Stu | ıdy design | .20 |
| 7. | PARTI | CIPANT SELECTION | .21 |
| | 7.1 Inc | lusion criteria | .22 |
| | 7.2 Ex | clusion criteria | . 22 |
| | 7.3 Est | timated sample size | .24 |
| ١ | | thdrawal criteria and loss to follow-up<br>Study protocol 4.0, 31 May 2021 | .24 |



| 7.5. | Security stop rules | 25 |
|---|---|---|
| 7.6 F | Recruitment period | 25 |
| 8. STUI | DY TREATMENT | 26 |
| 8.1 S | Study treatment | 26 |
| 8.2 E | Oosage | 26 |
| 8.3. I | Packaging and labelling | 26 |
| 8.4 T | reatment compliance | 26 |
| 8.5 C | Other treatments permitted and prohibited | 26 |
| 9. STUI | DY DEVELOPMENT AND PROCEDURES | 28 |
| 9.1 S | Study visits and procedures | 30 |
| 9.2 E | Biological samples | 34 |
| 10. EV | ALUATION CRITERIA: STUDY VARIABLES | 34 |
| 10.1 | Primary endpoint | 34 |
| 10.2 | Secondary endpoints | 34 |
| 10.3 | Bias control and limitations | 36 |
| 11 STU | DY SAFETY | 37 |
| 11.1 | Drug safety reference information | 37 |
| 11.2 | Definitions | 37 |
| 11.3 | Casualty evaluation | 39 |
| 11.4 | Intensity evaluation | 39 |
| 11.5 | Safety variables and parameters | 39 |
| 11.6 | Adverse events information | 39 |
| 11.7 | Pregnancy | 40 |
| 11.8 | Notification procedure of SAEs | 41 |
| 11.9 | Notification procedure of severe and unexpected adverse events (SUSAR) | 42 |
| VOLVE | R Study protocol 4.0, 31 May 2021 | |



| 12 | ? I | ETHICAL ISSUES | 43 |
|---|---|---|---|
| | 12.1 | General and particular rules for investigators | 43 |
| | 12.2 | Informed consent | 43 |
| | 12.3 | Safety and confidentiality procedures | 43 |
| | 12.4 | Insurance | 44 |
| 13 | 3 I | PRACTICAL CONSIDERATIONS | 44 |
| | 13.1 | Responsibilities of participants in the study | 44 |
| | 13.2 | Monitoring, auditing and inspection | 45 |
| | 13.3 | Study documentation | 45 |
| | 13.4 | Data management | 45 |
| | 13.5 | Publication conditions | 46 |
| | 13.6 | Procedure for the modifications of the protocol | 46 |
| | 13.7 | Ethics committee of research with medicines (CEIC) | 46 |
| 14 | | STATISTICAL ANALYSIS | 47 |
| | 14.1 | Sample size estimation | 47 |
| | 14.2 | Statistical analysis | 47 |
| 15 | . REF | ERENCES | 49 |
| A | PPEN | DIX 1. GUIDANCE ON PREGNANCY AND BREAST FEEDING | 53 |
| A | PPEN | DIX 2: RISK ASSESSMENT AND TOXICITY MANAGEMENT | 56 |
| | Risk / | Assessment | 56 |
| | Toxic | ity Management | 61 |
| A | PPEN | DIX 3: Liver Safety – Checklist for Drug Restart Approval or Refusal | 69 |
| A | PPEN | DIX 4: SERIOUS ADVERSE EVENT REPORT FORM | 70 |
| A | PPEN | DIX 5: PREGNANCY NOTIFICATION FORM | 72 |
| V | OLVEF | Study protocol 4.0. 31 May 2021 | |



| APPENDIX 6: PREGNANCY FOLLOW-UP FORM | 74 |
|-------------------------------------------------------------|----|
| APPENDIX 7: LIVER EVENTS FORM | 76 |
| APPENDIX 8: LIVER EVENTS BIOPSY FORM | 84 |
| APPENDIX 9: POSSIBLE SUICIDALITY-RELATED ADVERSE EVENT FORM | 91 |
| APPENDIX 10. LIVER IMAGING RECORD | 97 |



#### 3. GENERAL INFORMATION

## 3.1 Study identification

Clinical study title: Virologic Outcomes of Lamivudine/Dolutegravir in Virologically suppressed subjects with Expected or confirmed Resistance to Lamivudine (VOLVER study).

### 3.2 Type of clinical study

Phase IIa, open-label, single arm, multicentric study. Follow up: 96 weeks.

# 3.2 Study drug description

Dovato® (Dolutegravir 50 mg/Lamivudine 300 mg film-coated tablet):

Route of administration: oral.

Dose: Dolutegravir 50 mg/Lamivudine 300 mg/day.

Dosage: one 50 mg/300 mg film-coated tablet once daily.

Intervention: change of current antiretroviral treatment to DTG 50 mg/3TC 300 mg QD.

### 3.3 Principal investigators

Dr. José Ramón Arribas López

La Paz University Hospital.

Internal Medicine Department. Infectious Diseases Unit.

Paseo de la Castellana, 261. CP 28046 – Madrid

e-mail: joser.arribas@salud.madrid.org

#### Dr. Federico Pulido

Centro de Actividades Ambulatorias 2ª Planta Bloque D.

12 de Octubre University Hospital.

Av. Cordoba s/n. 28041-Madrid

e-mail: federico.pulido@salud.madrid.org

#### 3.4 Collaborating centres

Multicentre study, to be conducted at 17 healthcare centres in Spain. The listing of all investigators and sites will be attached in a separate document.

F S G
FUNDACIÓN
SEIMC-GESIDA

**GESIDA 11820** 

#### 3.5 Monitor identification

Fundación SEIMC-GESIDA.

C/ Agustín de Betancourt, 13-Entreplanta.

Tel: +34 91 556 80 25

Fax: +34 91 554 22 83

email: secretaria@f-sg.org

#### 3.6 Ethics committee of reference identification

Hospital La Paz Research Ethics Committee (Comité Ético de Investigación Clínica, CEIC).

Paseo de la Castellana, 261, 28046 Madrid.

e-mail: ceic.hulp.@salud.madrid.org

# 3.7 Expected duration

After obtaining the approval of the study by La Paz Research Ethics Committee (Comité Ético de Investigación Clínica) and by the Spanish Agency for Medicines and Health Products (Agencia Española del Medicamento, AEMPS), it is intended to carry out the study according to the following work plan:

- Duration of the participant selection period: 9 months.
- ii. Duration of the follow-up period: 96 weeks.
- iii. Data analysis and preparation of the final report: 6 months.

#### 4. BACKGROUND AND JUSTIFICATION

DTG/3TC is a dual regimen combination recommended for both naïve and suppressed persons with HIV-1 infection<sup>8</sup>. With the advent of DTG/3TC single tablet, a massive roll out of this antiretroviral therapy combination could be expected. Yet, data in treatment-experienced persons with past VF or resistances is currently insufficient to guarantee the robust benefits that DTG/3TC has already proved in large multicentric studies including naïve and suppressed persons without past resistances<sup>2,9</sup>.

3TC resistance-associated mutations are frequent in persons with past VF, with prevalence ranging from 34 to 96% depending on the setting, and the 2019 WHO HIV drug resistance report listing the M184V mutation as the most frequent mutation



associated with acquired NRTI drug resistance <sup>10–12</sup>. A retrospective study analysing 32,440 retrotranscriptase (RT) sequences of treatment-experienced persons found that about one third had codon 184 substitutions<sup>13</sup>. However, our group has demonstrated that 3TC resistance-associated mutations may not be detectable overtime as proviral DNA in suppressed persons detected only 26.9% of past M184V/I mutations<sup>14</sup>. At present, it is still unknown if proviral DNA genotyping in virologically suppressed patients can predict the efficacy of a given treatment, as this assay may not detect all previously existing drug-resistance mutations<sup>15–17</sup>. The importance of detecting minority resistant populations in proviral DNA is even more questionable since a high proportion of archived HIV is non replicating<sup>18,19</sup>. In addition, there is currently very little information on the relevance of those minority resistant populations detected by NGS, but not through proviral DNA population sequencing. To our knowledge, no study has prospectively investigated the dynamics of archived minority resistant variants in the presence of the drug to which they are theoretically resistant.

Studies in virologically failing patients have shown that 3TC retains antiviral efficacy despite evidence of 3TC resistance-associated mutations<sup>20–22</sup>. The MOBIDIP study was the first trial evaluating a dual regimen including 3TC for maintenance of HIV suppression in persons with history of 3TC resistance-associated mutations. In said study, 265 virologically suppressed participants- 96% of whom had a historical genotype detecting the M184V mutation- were randomized to either boosted protease inhibitor monotherapy or to 3TC plus boosted protease inhibitor. The study was prematurely discontinued after 48 weeks because the proportion of VF with boosted protease inhibitor monotherapy was significantly higher compared to 3TC plus boosted protease inhibitor (difference between groups 21.8%)<sup>11</sup>. Considering these results and in the context of past 3TC resistance, it is reasonable to contemplate that combining 3TC to another drug with a high genetic barrier such as DTG would also succeed in maintaining virologic suppression.

Reintroducing 3TC paired with DTG has shown promising results as maintenance therapy in persons with past 3TC resistance. The current scarce evidence for this strategy comes mostly from retrospective cohort analysis, a small number of participants from the DOLULAM study and four participants from the TANGO study who were found



to have the M184V mutation in proviral DNA at baseline and remained with virologic suppression through 48 weeks<sup>3–5,23</sup>.

The only study prospectively evaluating the efficacy of DTG/3TC in suppressed persons with past 3TC resistance is our pilot study ART-PRO<sup>6</sup>, where we hypothesized that this combination would be effective in maintaining virologic control in integrase naïve persons if 3TC resistance-associated mutations were not detected on baseline proviral DNA Sanger sequencing. In our study, 18/21 persons with past M184V/I mutations, not detected at baseline through proviral DNA Sanger sequencing, were switched to DTG/3TC and have maintained virologic control for 96 weeks without any case of VF<sup>7</sup>. The three participants that did not reach week 96 were discontinued due to a DTGrelated insomnia and two protocol violations, where two participants included in the study had baseline M184V mutation and thus were prematurely removed from the study at week 12, despite sustaining undetectable VL (<50 copies/mL). Interestingly, archived 3TC-resistance associated mutations were detected at baseline through NGS over the 5% threshold in more than half of participants with past 3TC resistance, without any detrimental effect on viral control. Although showing promising results, ART-PRO study's generalizability is limited due to the small size and the exclusion of participants exposed to integrase inhibitors.

Reusing 3TC in persons with past resistance combined with DTG would not only open the possibility to recycle 3TC but would also allow access to a simplified regimen endorsed by guidelines in participants who, owing to previous VF, are frequently excluded from clinical studies and treated with complex antiretroviral combinations that may include high pill burden or risk of toxicity. Therefore, we believe it is reasonable to perform a fully powered study designed to confirm the initial favourable results of our pilot study ART-PRO.

#### 5. HYPOTHESIS AND OBJECTIVES

#### 5.1 Hypothesis

Our hypothesis is that therapy with DTG/3TC would be able to maintain viral control in HIV infected participants with prior history of 3TC resistance but without evidence of M184V/I resistance mutation in provinal DNA population sequencing at baseline. We



also hypothesize that archived minority 3TC resistance associated mutations detected by next-generation (NGS) sequencing prior to the switch would not have a significant impact on the efficacy of DTG/3TC.

# 5.2 Objectives

| Primary objective | Primary endpoint |
|---|---|
| To assess the efficacy of a switch to DTG/3TC for maintenance of virologic suppression at 48 weeks in persons with past confirmed or suspected 3TC resistance, when proviral DNA population sequencing does not detect 3TC resistance-associated mutations at baseline. | Proportion of virologic failure (VF) defined as HIV-1 RNA viral load (VL) ≥50 copies per mL at 48 weeks (in the intention-to-treat-exposed population (ITT-e) using the US Food and Drug Administration (FDA) snapshot algorithm). |
| Secondary objectives | Secondary endpoints |
| To evaluate other estimations of virological control at weeks 48 and 96. | <ul> <li>Proportion of VF (≥50 copies/mL) at week 96, ITT-e, FDA snapshot.</li> <li>Proportion of VF (≥50 copies/mL) at week 48 and 96, per protocol population (PP), FDA snapshot.</li> <li>Proportion of VF (≥200 copies/mL) at week 48 and 96, ITT-e and PP population, FDA snapshot.</li> <li>Proportion of Confirmed Virologic Withdrawal ([CVW]: A VL≥ 50 copies/mL followed by a VL≥ 200 copies/mL in retest) at weeks 48 and 96, ITT-e and PP population, FDA snapshot.</li> <li>Proportion of Precautionary Virologic Withdrawal ([PVW]: three consecutive VL between 50- 200 copies/mL) at weeks 48 and 96, ITT-e and PP population, FDA snapshot.</li> <li>Proportion of participants with VL&lt;50 copies/mL week 48 and 96, ITT-e and per</li> </ul> |



| | protocol population, FDA snapshot. |
|---|---|
| To assess viral resistance in persons experiencing VF. | - Incidence of VF with drug resistance |
| | associated mutations. |
| | - Describe number and type of resistance- |
| | associated mutations in VF |
| | <ul> <li>Analysis of factors associated to VF (i.e time to VF).</li> </ul> |
| | - Proportion of VF in pre-specified |
| | subgroups: |
| To evaluate factors associated with VF. | - Confirmed historical M184V/I vs No |
| | resistance mutations |
| | - INSTI exposure vs No prior INSTI |
| | exposure |
| | - Time virologically suppressed |
| | - Time on 3TC/FTC |
| | - Proportion of participants with VF with |
| | baseline 3TC or INSTI resistance-<br>associated mutations detected at<br>baseline by NGS with 1, 5, and 20% |
| To assess the impact of baseline archived | |
| minority 3TC resistance-associated mutations | |
| in viral control (in cases of VF and transient | threshold. |
| viral rebounds [VL≥50copies/mL preceded | - Proportion of participants with transient |
| and followed by VL<50 copies/mL]). | viral rebounds with baseline 3TC or INSTI |
| | resistance- associated mutations |
| | detected at baseline by NGS with 1, 5, |
| | and 20% threshold. |
| To evaluate the dynamics of archived minority | Type and frequency of resistance mutations |
| 3TC resistance-associated mutations after | (RT and integrase) in proviral DNA measured |
| switching to DTG/3TC at 96 weeks. | by NGS at baseline and week 96. |
| To evaluate the immune effects of switch to | Change from Baseline in CD4+ cell count and |
| DTG/3TC | in CD4+/CD8+ cell counts ratio at weeks 48 |
| | and 96 |
| To evaluate the safety and tolerability of | - Incidence and severity of AEs and laboratory abnormalities through week 48 |
| DTG/3TC in this study | and 96. |
| | and 96. |



| • | Proportion of subjects who discontinue |
|---|----------------------------------------|
| | treatment due to AEs through weeks 48 |
| | and 96. |

#### 6. TYPE OF CLINICAL STUDY AND DESIGN

### 6.1 Clinical study phase

Phase IIa study.

### 6.2 Study design

Open, single-arm, multicentric study evaluating the efficacy and safety of DTG/3TC as maintenance therapy for HIV-1 virologic suppression in persons with historical 3TC resistance.

The study consists of a Screening phase (maximum 60 days prior to day 1), and a Switch phase (day 1).

The study will screen for adult participants with HIV infection with history of confirmed or suspected resistance to 3TC receiving stable ART for at least 12 weeks and virologically supressed for at least one year prior to the study entry. Participants who provide informed consent and meet inclusion criteria will be screened in order to enrol 120 subjects.

On day 1 all participants who meet study entry criteria will be switched to DTG/3TC. There will be two groups: one group with confirmed historical 3TC resistance mutation, that is, with the M184V/I in an historical RNA Sanger genotype (minimum 30%-50% of the study population), and another group with suspicion of 3TC resistance based on clinical and virological history. No participant with M184V/I or K65R detected in screening proviral DNA population sequencing will be allowed to enter the study. Participants will attend study centres at screening, baseline, weeks 4, 12, 24, 36, 48 (primary efficacy endpoint), 72 and 96 (secondary efficacy endpoint, end-of-study visit). Primary endpoint is proportion of virologic failure at 48 weeks, following the FDA snapshot algorithm, ITT-

<sup>\*</sup>Intention- to -treat-exposed (ITT-e) includes all participants receiving at least one dose of DTG/3TC.

<sup>\*\*</sup>Per protocol (PP) analysis excludes participants with protocol violations, lost to followup and those with low adherence (adherence at or below the 2.5th percentile of those in the study).



e analysis. There will be a safety analysis at week 24 and also a "stopping rule" throughout the study, whereby if two cases of confirmed (CVW) or precautionary virologic withdrawal (PVW) occur with INSTI resistance at any timepoint, the study will be terminated (see section 7.4 for definitions for CVW and PVW). Procedures described in this protocol will be performed at each visit, including blood sampling for hemogram, biochemistry, HIV viral load and CD4 count. At screening and week 96, proviral DNA NGS will be performed. RNA sanger genotype and proviral DNA NGS will be performed in all cases of CVW and PVW.

Overall study design:



This study will be conducted in compliance with the protocol, Good Clinical Practice, and all applicable regulatory requirements.

#### 7. PARTICIPANT SELECTION

Subjects will be offered to participate in the study on the basis of the following eligibility criteria.



#### 7.1 Inclusion criteria

- a. Adults (≥ 18 years old) with HIV-1 infection able to understand and give informed written consent.
- b. Stable ART in the 12 weeks prior to study entry.
  - Only switch for tolerability/convenience/access reasons to generic drugs or switch from ritonavir to cobicistat or TDF to TAF would be allowed in the 12-week window and as long as the components of the regimen are unchanged.
- c. Viral load <50 copies/mL at screening and in the year prior to study entry.
  - A blip (50-500 copies/mL) would be allowed within 48 weeks prior to inclusion in the study, if preceded and followed by an undetectable VL determination (HIV-RNA <50 copies/mL).</li>
- d. CD4<sup>+</sup> count > 200 cells/μL at screening.
- e. History of 3TC resistance: either *confirmed historical 3TC resistance* (historical RNA Sanger or RNA NGS>20% threshold genotype with M184V/I mutation) OR *suspected historical 3TC resistance*.
  - Suspicion of past 3TC resistance is defined as <u>any</u> of the following:
    - i. Previous treatment with only 2 NRTIs (1 of them being emtricitabine or 3TC [XTC]).
    - ii. Two consecutive VL > 200 copies/mL while on treatment including XTC.
    - iii. One VL > 200 copies/mL while on treatment including XTC <u>PLUS</u> change of ART as consequence of that elevated VL.

#### 7.2 Exclusion criteria

- a. Participants with M184V/I or K65R in screening visit proviral DNA Sanger genotype.
- b. Prior virologic failure (VF) under integrase inhibitor (INSTI)- based regimen.
   defined as two consecutive VL > 200 copies/mL while receiving INSTI regardless of genotypic test results
- c. INSTI resistance mutations in historical RNA genotype



- d. Documented resistance to DRV defined as the presence of a combination of mutations scored with at least 15 points in the Stanford University HIV Drug Resistance Database.
- e. Positive Surface Hepatitis B Ag (HBAgS) OR negative HBAgS and negative hepatitis B surface antibody (anti-HBs) with positive anti-core antibody (anti-HBc) and positive HBV DNA.
- f. Pregnant, breastfeeding women, women with a positive pregnancy test at the time of screening, sexually active fertile women wishing to conceive or unwilling to commit to contraceptive methods (see Appendix 1 for the accepted list of the highly effective methods for avoiding pregnancy), for the duration of the study and until 4 weeks after the last dose of study medication. All women are considered fertile unless they have undergone a sterilizing surgery or are over the age of 50 with spontaneous amenorrhea for over 12 months prior to study entry.
- g. Patients with active opportunistic infections or cancer requiring intravenous treatment and/or chemotherapy at screening.
- h. Any comorbidities or treatment with experimental drugs that according to the investigator could bias study results or entail additional risks for the participant.
- i. Participants receiving other medications that according to study drug label are contraindicated.
- j. Severe hepatic impairment (Class C) as determined by Child-Pugh classification.
- k. Alanine aminotransferase (ALT) over 5 times the upper limit of normal (ULN) or ALT over 3xULN and bilirubin over 1.5xULN.
- Unstable liver disease (as defined by the presence of ascites, encephalopathy, coagulopathy, hypoalbuminemia, esophageal or gastric varices, or persistent jaundice), cirrhosis, known biliary abnormalities (apart from hyperbilirubinemia or jaundice due to Gilbert's syndrome or asymptomatic gallstones);
- m. Creatinine clearance of <30 mL/min/1.73m<sup>2</sup> via CKD-EPI method.
- n. Any verified Grade 4 laboratory abnormality that to the investigators criteria would affect the safety of the participant if included in the study.
- o. History or presence of allergy to dolutegravir or lamivudine.



### 7.3 Estimated sample size

In previous studies of switch to DTG/3TC the rate of VF at week 48 has been  $0.7\%^{24}$ . With 120 participants recruited, and considering the same proportion of VF, we could rule out differences in the proportion of VF > 4% with a binomial estimation of the 95% confidence interval (power 80%, alpha 5% bilateral).

There will be two groups of participants: one with *confirmed* history of 3TC resistance based on historical RNA genotype and another one with *suspected* 3TC resistance based on clinical and virologic history. The group with confirmed 3TC resistance will comprise at least between 30-50% of the estimated sample size.

### 7.4 Withdrawal criteria and loss to follow-up

In accordance with the current revision of the Declaration of Helsinki (Fortaleza, Brazil October 2013)<sup>25</sup> and with the applicable regulations, a participant has the right to withdraw from the study at any time and for any reason, without prejudice to the medical care provided by his doctor and /or referral centre in the future. A participant may be withdrawn from the study in the following scenarios:

- Participant withdraws consent.
- For safety reasons. In particular, subjects will be withdrawn from the study if any of the following occur:
  - i. If adverse events (AEs) appear and, due to their type or severity,
    cause the participant not to remain in the study. See Appendix
    2: Toxicity Management.
  - ii. Pregnancy.
  - iii. Subject is incorrectly included in the study based on exclusionary screening proviral DNA lamivudine resistance or any other protocol exclusion criteria.
  - iv. Subject meets criteria for Confirmed Virologic Withdrawal or Precautionary Virologic Withdrawal.
    - Confirmed Virologic Withdrawal (CVW):
      - A VL≥ 50 copies/mL followed by a VL≥ 200 copies/mL in re-test 2-4 weeks apart.
    - Precautionary Virologic Withdrawal (PVW)



- Three consecutive VL 50-200 copies/mL (each VL separated 2-4 weeks).
- At investigator discretion based on good clinical practice guidelines and clinical judgement deeming the participant ineligible to continue the study.
- Transfer to another hospital that is not a participating centre in the study.
- Loss to follow-up.
- The participant is not willing to comply with the procedures required in the protocol.

The causes leading to withdrawal from the study will be clearly recorded in the Clinical Research Document (CRD). A specific Withdrawal Visit will be scheduled to detail the participant's evolution, date of treatment discontinuation and new prescribed therapy (if applicable). If any ongoing AE is present at the time of Withdrawal Visit, the participant will be followed until its resolution or stabilization.

Participants discharged from the study will return to usual care according to the local guidelines and clinical practice.

Withdrawn participants may be replaced to achieve the estimated sample size, provided the stopping rule does not apply.

#### 7.5. Security stop rules

Study will be terminated at any timepoint if two cases of CVW or PVW with development of INSTI resistance occur.

A security analysis will take place at week 24. Study will be prematurely discontinued if less than 80% participants in the per protocol population have VL<50 copies/mL (FDA-Snapshot algorithm).

#### 7.6 Recruitment period

Study recruitment period is estimated in nine months, alternatively, until sample size is achieved.

A 60-day window is established between screening visit and day 1 visit.

If CD4<sup>+</sup> count or VL inclusion criteria are not met on first screening visit, one re-screening visit within 4 weeks would be allowed per participant. Re-screening visit will only be

F S G
FUNDACIÓN
SEIMC-GESIDA

**GESIDA 11820** 

performed if deemed appropriate by Medical Monitor and the investigator after detailed review of clinical history and mitigating factors.

#### 8. STUDY TREATMENT

# 8.1 Study treatment

DTG/3TC (Dovato®).

#### 8.2 Dosage

Dovato® (Dolutegravir 50 mg/Lamivudine 300 mg film-coated tablet):

Route of administration: oral.

Dose: Dolutegravir 50 mg/Lamivudine 300 mg/day.

Dosage: one 50 mg/300 mg film coated-tablet once daily.

Intervention: change of current antiretroviral treatment by DTG 50 mg/3TC 300 mg QD.

### 8.3. Packaging and labelling

Dovato® will be supplied by the hospital Pharmacy Department of each participating site for the treatment of their respective patients, dispensed in a controlled fashion and according to hospital directives.

The containers of Dovato® will be provided by the study Sponsor and the labelling for the study will be done by an outside agent in accordance with current national legislation.

# 8.4 Treatment compliance

Treatment adherence will be assessed by active questioning at study visit plus pill count, every visit from week 4 through week 96/end of study. Study drug will be labelled according to subject identification code, visit number and date. At every visit, the remaining medication will be returned by the participant to be counted and collected, and new medication will be assigned.

#### 8.5 Other treatments permitted and prohibited

At study initiation, all concomitant medications will be recorded in the CRD and checked for potential drug-drug interactions at "https://www.hiv-druginteractions.org/checker".



Thereafter, all changes in medication will be detailed in the CRD. Additionally, all diagnostic, therapeutic or surgical procedures performed during the study period will be recorded, including date, indication, description of the procedure and clinical findings.

# Prohibited drugs

The following medications or their equivalents can cause a decrease in the concentration of DTG and therefore should not be administered simultaneously with DTG.

- Carbamazepine
- Oxcarbamazepine
- Phenobarbital
- Phenytoin
- Rifampin or rifapentine
- St. John's wort

DTG/3TC is contraindicated with co-administration of medicinal products with narrow therapeutic windows, that are substrates of organic cation transporter (OCT2), including but not limited to fampridine (also known as dalfampridine). Co-administration has the potential to cause seizures due to increased fampridine plasma concentration.

NOTE: DTG should be administered 2 hours before or 6 hours after medicines with divalent cations (Ca<sup>++</sup>, Fe<sup>++</sup>), multiple vitamin supplements or antacids containing aluminium or magnesium salts.

All treatments considered experimental will be prohibited during the study.



# 9. STUDY DEVELOPMENT AND PROCEDURES

| Visit | V0 | V1 | V2 | V3 | V4 | V5 | V6 | V7 | V8 | V9 |
|---|---|---|---|---|---|---|---|---|---|---|
| Week | Screening | D1<br>(Basal<br>visit) | W4<br>(±2<br>days) | <b>W12</b> (± 4 days) | <b>W24</b> (± 6 days) | <b>W36</b> (±6 days) | <b>W48</b><br>(± 6<br>weeks) | <b>W72</b> (±8 days) | W96<br>(±6<br>weeks) | Follow<br>up |
| Informed Consent | x | | | | | | | | | |
| Inclusion and exclusion criteria | х | х | | | | | | | | |
| Screening visit assessments | х | | | | | | | | | |
| Physical Exam <sup>†</sup> | × | x | x | x | x | x | x | x | x | |
| Vital signs and BMI | х | х | х | х | х | х | х | х | х | |
| Laboratory assessment<br>(hemogram, chemistry<br>including renal and hepatic<br>function tests) | x | х | х | х | х | х | x | х | x | |
| Pregnancy test (if applicable), blood or urine | х | х | х | х | х | х | х | х | х | |
| Quantitative plasma HIV-1<br>RNA | х | х | х | x | х | х | x | х | x | |
| CD4 <sup>+</sup> and CD8 <sup>+</sup> count cells/µL | х | х | х | х | х | х | х | х | х | |
| PBMC proviral DNA RT Sanger sequencing | x | | | | | | | | | |



| PMBC Proviral DNA RT,<br>PR and INSTI NGS | х | | | | | | | | х | |
|---|---|---|---|---|---|---|---|---|---|---|
| Dispense study treatment | | x | x | x | x | х | х | х | | |
| Study treatment pill count | | | х | х | х | х | х | х | х | |
| Concomitant Medication review | х | х | х | х | х | х | Х | х | Х | х |
| Adverse Events | Х | х | х | х | х | х | х | х | х | х |

Table 1. Evaluation calendar per visit.

A 60-day window is allowed between screening visit and day 1. Re-screening would only be allowed under special circumstances and careful evaluation by Medical Monitor and investigator (see section 7.6)

For the endpoint visits (week 48 and 96) a ±6-week window is allowed.

Withdrawal visit will be performed if any subject prematurely discontinues the study, see specific assessments in section 9.1

All serious adverse events will be reported from the moment the written informed consent is signed (see section 11 [Study safety]).

A Follow-up visit will be scheduled 28 days after the last dose of study medication to monitor and report any ongoing adverse event or laboratory abnormality considered to be potentially harmful for the participant.

<sup>&</sup>lt;sup>†</sup> Physical exam will be performed symptom-orientated from day 1 (V1) onwards.



### 9.1 Study visits and procedures

The study will be offered to participants that meet all the inclusion criteria and none of the exclusion criteria. There will be a total of 10 visits (screening, day 1, week 4, week 12, week 24, week 36, week 48, week 72, week 96 and a follow-up visit).

#### Screening visit:

Participants will receive the information relative to proceedings and study visits. If they agree to participate in the study, written informed consent should be signed before any procedure is performed. Screening assessments include:

- Review of inclusion and exclusion criteria.
- Demographic data: age, sex, race, country of origin
- HIV infection data: HIV subtype, mode of transmission, HIV + diagnosis date, nadir CD4<sup>+</sup>, CDC stage, presence of previous AIDS diagnosis, HIV associated conditions, ART duration, time with VL <50 copies/ mL (excluding one blip [50-500 copies/mL preceded and followed by a VL<50 copies/mL] in the year prior to study entry), previous antiretroviral treatments (number, type, reasons for change, date of change), resistance studies (resistance mutations detected in historical genotypic population studies, date of the genotypic study, viral load detected during the genotypic study).</p>
- General medical history: previous illnesses, active diseases, active treatments, tobacco, alcohol and drug habits.
- Physical exam including weight, height, BMI, blood pressure and heart rate.
- Adverse events.
- Laboratory assessments will include:
  - Hemogram
  - Chemistry: liver function tests, renal function tests, fasting lipids, glucose.
  - o Pregnancy test in women of childbearing potential (blood or urine



sample)

- AgHBs, antiHBc, antiHBs and HBV DNA in those with isolated antiHBc (if not performed in the 12 months prior to screening visit).
- CD4<sup>+</sup> and CD8<sup>+</sup> count.
- Viral load (quantitative plasma HIV-1 RNA)
- PBMC DNA Sanger sequencing (RT): using Big Dye Terminator (Applied Biosystem), and the Stanford HIVDB algorithm to interpret resistance mutations
  - PBMC proviral DNA NGS sequencing (integrase, protease and RT) sample will be saved to be performed retrospectively if participant continues to switch phase. For NGS, HIV-1 DNA will be extracted from PBMCs using the QIAamp® DNA blood minikit (Qiagen, Hiden, Germany) and a 3385 bp pol gene fragment will be amplified by nested PCR as described elsewhere<sup>26</sup>. NGS will be performed with Illumina in a Miseq instrument (Illumina, San Diego, CA, USA). Sequences wil be preprocessed with Prinseq-lite (http://prinseq.sourceforge.net/) and FLASH (http://www.cbcb.umd.edu/software/flash) programs<sup>27,28</sup>. The resulting aligned reads will be analyzed for HIV-1 drug resistance testing with PaSeq software (https://paseq.org/). The 1% threshold is for resistance interpretation. Baseline samples with 3TC or integrase resistance-associated mutations detected through NGS will undergo 2.0 hypermutation analysis with Hypermut software (https://www.hiv.lanl.gov/content/sequence/hypermut/hypermut.html).

# <u>Day 1:</u>

- Review of inclusion and exclusion criteria.
- Concomitant medication.
- Adverse events.
- Physical exam including weight, height, BMI, blood pressure and heart rate.



- Switch to study treatment: DTG/3TC 50/300 mg once daily.
- Laboratory assessments will include:
  - Hemogram.
  - Chemistry: liver function tests, renal function tests, fasting lipids, glucose.
  - CD4<sup>+</sup> and CD8<sup>+</sup> count.
  - Viral load (quantitative plasma HIV-1 RNA).
  - Pregnancy test if women of childbearing potential (blood or urine sample)

# Visits week 4 to week 96:

- Concomitant medication.
- Adverse events.
- Physical exam including weight, height, BMI, blood pressure and heart rate.
- The remaining study medication will be counted and collected, and new medication will be dispensed.
- Laboratory assessments will include:
  - Hemogram.
  - Chemistry: liver function tests, renal function tests, fasting lipids, glucose.
  - CD4<sup>+</sup> and CD8<sup>+</sup> count.
  - Viral load (quantitative plasma HIV-1 RNA).
  - Pregnancy test if women of childbearing potential (blood or urine sample).
- Week 96 additional assessments:
  - PBMC proviral DNA NGS sequencing (integrase, PR and RT)



In the event of a VL≥ 50 copies/mL at any time point between day 1 and week 96, a visit will be scheduled within 2-4 weeks to perform a VL re-test.

A Follow-up visit will be scheduled 28 days after the last dose of study medication to monitor and report any ongoing adverse event and concomitant medication or laboratory abnormality considered to be potentially harmful for the participant.

Investigators are allowed to perform additional assessments and procedures following local guidelines and clinical criteria (i.e vaccination, sexually transmitted infection screening), as long as they are not judged to interfere with study proceedings and are registered with detail in the medical history.

After week 96 study visit, the investigator is responsible for ensuring that the participants have continued access to antiretroviral treatment.

### Withdrawal Study Visit:

If at any given point the participant is prematurely discontinued from the study, for any of the specified reasons in section 7.4 a Withdrawal Study Visit will be performed and registered in the CRD. This visit will include:

- Concomitant medication.
- Adverse events.
- Physical exam including weight, height, BMI, blood pressure and heart rate.
- Pregnancy test if women of childbearing potential (blood or urine sample).
- The remaining study medication will be counted and collected.
- Laboratory assessments will include:
  - Hemogram.
  - Chemistry: liver function tests, renal function tests, fasting lipids, glucose.
  - CD4<sup>+</sup> and CD8<sup>+</sup> count.
  - Viral load (quantitative plasma HIV-1 RNA).



If <u>CVW or PVW</u> occur, resistance test (RNA Sanger sequencing, integrase, PR and RT, ViroSeq HIV-1 Genotyping System (Abbott Molecular, Spain) and PBMC proviral DNA NGS sequencing (integrase, PR and RT) will be performed.

# 9.2 Biological samples

All genotyping analysis will be centralized in 12 de Octubre University Hospital:

- a. Proviral DNA population sequencing (Sanger, RT) and NGS (RT, PR, integrase)
  - i. Sample: PBMC (10 mL blood, CPT tube).
  - ii. Screening visit and also week 96 for NGS.
- RNA population sequencing (Sanger, RT, PR, integrase) and PBMC proviral DNA
   NGS sequencing (integrase, PR and RT) in the event of CVW or PVW:
  - Samples: Peripheral blood (10 mL blood, CPT tube) and PBMC (10 mL blood, EDTA tube).
  - ii. Any timepoint throughout the study.

#### 10. EVALUATION CRITERIA: STUDY VARIABLES

## 10.1 Primary endpoint

Proportion of virologic failure defined as HIV-1 RNA viral load ≥50 copies per mL at 48 weeks, ITT-e population, using the US Food and Drug Administration (FDA) snapshot algorithm).

ITT-e includes all participants receiving at least one dose of DTG/3TC.

#### 10.2 Secondary endpoints

- a. Proportion of VF (≥50 copies/mL) at week 96, ITT-e, FDA snapshot.
- b. Proportion of VF (≥50 copies/mL) at week 48 and 96, per protocol population, FDA snapshot. Per protocol population excludes participants with protocol violations, lost to follow-up and those with low adherence (adherence at or below the 2.5th percentile of those in the study).
- c. Proportion of VF (≥200 copies/mL) at week 48 and 96, ITT-e and PP population, FDA



snapshot.

- d. Proportion of CVW at weeks 48 and 96, ITT-e and PP population, FDA snapshot.
- e. Proportion of PVW at weeks 48 and 96, ITT-e and PP population, FDA snapshot.
- f. Proportion of participants with VL<50 copies/mL week 48 and 96, ITT-e and PP, FDA snapshot.
- g. Incidence of VF with drug resistance associated mutations.
- h. Description of number and type of resistance-associated mutations in VF.
- i. Analysis of factors associated to VF (i.e time to VF).
- j. Proportion of VF in pre-specified subgroups:
  - Confirmed historical M184V/I vs No documented resistance mutations.
  - INSTI exposure vs No prior INSTI exposure.
  - Time virologically suppressed
  - Time on 3TC/FTC.
- k. Proportion of participants with VF with baseline 3TC or INSTI resistance- associated mutations detected at baseline by NGS with 1, 5, and 20% threshold.
- Proportion of participants with transient viral rebounds with baseline 3TC or INSTI resistance- associated mutations detected at baseline by NGS with 1, 5, and 20% threshold.
- m. Type and frequency of resistance mutations (RT and integrase) in proviral DNA measured by NGS at baseline and week 96.
- n. Change from Baseline in CD4<sup>+</sup> cell count and in CD4<sup>+</sup>/CD8<sup>+</sup> cell counts ratio at weeks 48 and 96.
- o. Incidence and severity of AEs and laboratory abnormalities through week 48 and 96.
- Proportion of subjects who discontinue treatment due to AEs through weeks 48 and
   96.
- q. Descriptive demographic and clinical variables:
  - Demographic data: age, sex, race, country of origin
  - HIV infection data: HIV subtype, mode of transmission, HIV + diagnosis date, nadir CD4<sup>+</sup>, CDC stage, presence of previous AIDS diagnosis, HIV associated conditions, ART duration, time with viral load <50 copies/mL (excluding one blip [50-500 copies/mL preceded and followed by a VL<50 copies/mL] in the year prior to study entry), previous antiretroviral treatments (number, type, reasons



for change, date of change), resistance studies (resistance mutations detected in historical genotypic population studies, date of the genotypic study, viral load detected during the genotypic study, time since the virological failure or interruption of antiretroviral treatment and the completion of the genotypic study.

- General medical history: previous illnesses, active diseases, active treatments, tobacco, alcohol and drug habits.
- Physical exam including weight, height, BMI, blood pressure and heart rate.
- Laboratory assessment variables: Haemoglobin, leukocytes, lymphocytes, neutrophils, CD4<sup>+</sup> and CD8<sup>+</sup>, GOT, GPT, GGT, Bilirubin, Creatinine, Ions, total cholesterol, HDL, LDL, triglycerides, glucose.

#### 10.3 Bias control and limitations

The absence of 3TC resistance mutations in the population genotype of proviral DNA Sanger does not guarantee the success of DTG/3TC treatment. However, based on the results from our pilot study ART-PRO<sup>29</sup>, we believe that this is a reasonable working hypothesis. If any case of VF occurred, proviral DNA RT+ INSTI NGS for retrospective analysis will allow to detect if any archived resistance minority variants were present at baseline and could therefore be the cause of failure.

Proviral HIV analysis could be limited by the number of latently infected CD4 lymphocytes present in the sample, so PBMCs will be used to ensure maximum resistance detection capacity.

Objective primary and secondary endpoints will allow to reduce the potential bias associated with the open label design of the study.


#### 11 STUDY SAFETY

#### 11.1 Drug safety reference information

In this study, the reference safety information will be the European Medicine Agency Dovato® product information<sup>30</sup>.

#### 11.2 Definitions

#### Adverse event (AE):

Any medical event presented by a clinical research subject to whom a pharmaceutical product has been administered and does not necessarily have to have a causal relationship with said treatment.

The following will be registered as an AE:

- Significant or unexpected worsening of the condition to be treated during the study.
- Exacerbation of pre-existing chronic, intermittent or episodic diseases, including an increase in frequency and /or severity.
- A new condition detected or diagnosed after the administration of the product under investigation, even if it could have been present before study initiation.
- Suspicious clinical signs, symptoms or sequelae.
- Clinical signs, symptoms or sequelae of a suspected overdose of the medicinal product under investigation or concomitant medication.
- Obvious failure of the expected biological or pharmacological effect.
- Any medical reaction before, during or after the treatment resulting from the procedures specified in the protocol, such as those derived from sampling.
- Grade III-IV laboratory events, as classified by DAIDS toxicity scales<sup>31</sup>.

It will not be considered, and therefore not recorded as an AE:

- Medical or surgical procedures due to the course of the disease allowed in the clinical study.
- Situations leading to hospital admission for social or convenience reasons, VOLVER Study protocol 4.0, 31 May 2021



without any medical underlying reasons.

- Clinical signs, symptoms or sequelae of the study disease or its expected progression.

#### Serious adverse event (SAE):

Any medical event leading to:

- Death
- Life endangerment
- Hospital admission, prolongation of existing hospital admission
- Persisting or significant disability / incapacity, or results in a congenital anomaly or defect.
- All events of ALT ≥ 3xULN and bilirubin ≥ 2xULN (>35% direct bilirubin) or ALT ≥ 3xULN and INR>1.5 (if INR measured) which may indicate severe liver injury must be reported as a serious adverse event (excluding studies of hepatic impairment or cirrhosis).
- Events not included in the preceding paragraphs but that may endanger the
  participant or require intervention to prevent any of the abovementioned
  results. Examples of such events are intensive treatment in an emergency
  department or at home for an allergic bronchospasm; blood dyscrasias or
  seizures that do not lead to hospital admission, or the development of
  dependence or drug abuse.

For notification purposes, suspicions of AEs that are considered medically important will be treated as serious, even if they do not meet the above criteria, such as those that put the participant at risk or require intervention to prevent any of the abovementioned outcomes.

#### <u>Unexpected Serious Adverse Reaction (SUSAR):</u>

Any serious adverse event which nature, severity or consequences are not consistent with the available product information.



#### 11.3 Casualty evaluation

Investigators will assess casualty of the AE with the study medication according to the following definitions:

| Relatedness Rating | Definition |
|---|---|
| Related | An adverse event in which there is a reasonable possibility of a causal relationship to |
| | the use of the study drug. 'A reasonable possibility' is meant to convey that there are |
| | facts/evidence or arguments to suggest a causal relationship. Facts/evidence or |
| | arguments that may support 'a reasonable possibility' include, e.g. a temporal |
| | relationship, a pharmacologically-predicted event, or positive dechallenge or |
| | rechallenge. Confounding factors, such as concomitant medication, a concurrent |
| | illness, or relevant medical history, should also be considered. |
| Not Related | An adverse event which is not related to the use of the drug. |

#### 11.4 Intensity evaluation

The intensity of the AE will be graded following the DAIDS grading table for Severity of AEs<sup>31</sup>.

#### 11.5 Safety variables and parameters

To investigate AEs, investigators will enquiry at every visit for AEs. To avoid bias and to promote spontaneous report of AEs, questions addressed to participants will be open and are not to have a leading nature. Questions may be as:

- How are you?
- Have you presented any symptoms since the last visit?
- Have you needed evaluation by another healthcare professional?
- Have you visited any emergency department?
- Have you taken any other medications besides antiretroviral treatment since the last visit? If so, why?

#### 11.6 Adverse events information

All SAEs and AEs will be collected from the signing of the ICF until the follow-up visit.



All AEs occurring during the study, until the end of the follow-up period, whether or not they are attributed to the study medication, will be evaluated by the investigator and recorded in detail in the CRD. Data on the description of the AE, start and end date, severity/intensity, causality with the investigational drug product, evolution, outcome of the AE and measures adopted (treatments, additional complementary examinations) will be recorded, including those related to the investigational medication (eg, suspension). Regardless of the causal relationship with the study drug, all AE will be followed until resolution or until considered stable. The investigator is authorized to judge if the severity of the AE requires discontinuation of the treatment or participant withdrawal from the study. Participants may also voluntarily withdraw if they perceive an AE as not tolerable. A Follow-up visit will be scheduled 28 days after the last dose of study medication to monitor and report any ongoing adverse event or laboratory abnormality considered to be potentially harmful for the participant.

The outcome of the AE will be evaluated as follows:

- Resolved.
- Improved
- Unchanged.
- Worsening.
- Death.

Action taken by the investigators with regards to the study medication:

- None.
- Discontinuation.
- Interruption.
- Dose reduction.
- Delay in the beginning of treatment.

#### 11.7 Pregnancy

Female participants will be instructed to notify the investigator if they become pregnant at any time during the study.



Women of childbearing potential should be informed about the potential risk of neural tube disorders with DTG (see Appendix 1). These defects happen early in pregnancy, before women may know they are pregnant.

Women of childbearing age should use an appropriate contraceptive method for the duration of the study and up to 4 weeks after completion (see Appendix 1, Guidance on Pregnancy and Breast Feeding). The chosen contraceptive method will be documented in the subject's medical records. Women of childbearing potential will be informed of the potential risk of neural tube defects and will be counselled on avoiding pregnancy, safer sexual practices and the proper use of their chosen contraceptive methods.

A pregnancy test (blood or urine) will be performed at every study visit. Any pregnancy occurring within the study will result in immediate withdrawal from the study and discontinuation of study drug treatment.

Each pregnancy will be notified to the Medical Monitor as soon as it is known to the investigator. Information will be recorded on the appropriate form (see Appendix 5 and 6) and submitted to the Sponsor within 24 hours of of learning of a subject's pregnancy. All pregnancies should also be reported to ViiV Healthcare within 1 week, regardless of causality. Additionally, pregnancies will be registered in the AntiretroviralPregnancy Registry (www.apregistry.com).

Pregnancy should be followed to determine the outcome, including spontaneous or voluntary termination, birth details, and the presence or absence of any defect such as congenital anomaly or complications for the mother and / or newborn. Pregnancy results should also be recorded for female partners of a male participant who is participating in the study. If the outcome of pregnancy meets SAE criteria or if the newborn has a SAE, the procedures described for the notification of SAE will be followed. Spontaneus abortions must be reported as a SAE.

#### 11.8 Notification procedure of SAEs

Investigators should notify the sponsor or whoever assumes the tasks delegated by the sponsor within a maximum period of 24 hours after learning of the existence of a SAE, with an accompanying SAE notification form.

The investigator shall complete and sign the SAE report form (Appendix 6) and send it by fax:





#### 915542283

# Fundación SEIMC-GESIDA C/ Agustín de Betancourt nº 13, entreplanta Madrid 28003

and/or email to: pharmacovigilance@f-sg.org

SAEs associated with DTG/3TC should also be reported to ViiV Healthcare within 24 hours, regardless of casualty. The sponsor or whoever assumes the tasks delegated by the sponsor may request additional information from the investigator. The investigator will provide information to the sponsor or to those who assume the tasks delegated by the sponsor whenever requested and, in any case, when their initial evaluation changes in terms of severity or causality. The sponsor or whoever assumes the tasks delegated by the sponsor will keep a detailed record of all the SAEs communicated to them by the researchers.

#### 11.9 Notification procedure of severe and unexpected adverse events (SUSAR)

The sponsor or whoever assumes the tasks delegated by the sponsor, will notify all the suspicions of SUSAR according to the current regulations on clinical trials to the Spanish Agency of Medicine and Health Products (AEMPS), to the ethical committees (CEIC) and to the authorities of the Autonomous Community of Madrid within a maximum period of fifteen calendar days from the moment they are aware of their existence. When the SUSAR has caused the death of the participant or endangered his life, the notification will be made within a maximum period of seven calendar days from the moment in which it is known. The relevant information regarding subsequent events will be supplemented within eight days.

The minimum initial information for the notification of an adverse event must include the following:

- Adverse event and starting date.
- Initials, sex and age (or date of birth) of the participant.
- Information about the treatment received.

VOLVER Study protocol 4.0, 31 May 2021



- Name and address of the doctor notifying the AE.
- Causality relationship with the medication under study.

#### 12 ETHICAL ISSUES

#### 12.1 General and particular rules for investigators

Investigators will strictly adhere to the provisions of this protocol, fully completing the data collection notebook sheets.

The study will follow the prevailing recommendations for medical research involving human subjects, as reflected in the latest version of the Declaration of Helsinki and the current the applicable Spanish Legislation on Clinical Studies (RD 1090/2015, of December 4, which regulates clinical trials with medications).

#### 12.2 Informed consent

All participants will be informed before starting the study of the objectives, procedures, potential related inconveniences derived from said procedures, and the risks of the study. All subjects will receive a participant information sheet, along with the written informed consent that must be signed at screening visit before any procedure relating to the study is performed.

#### 12.3 Safety and confidentiality procedures

All information obtained from this study is considered confidential. The confidentiality of the personal and genetic data obtained will be protected, respecting at all times the basic ethical principles of research with biological samples, and as established by the applicable legislation (Regulation 2016/679 of the European Parliament and of the Council of 27 April 2016 on the protection of natural persons with regard to the processing of personal data and on the free movement of such data).

Participants may at any time exercise their right to access and modify their information, as established by the Spanish Organic Law for Personal Data Protection 3/2018 and the European General Data Protection Regulation 2016/679.



In case of considering the participation in a new study, with a different objective to that indicated in the information sheet, the participant will be informed and new consent and permission to use the samples will be requested. Biological samples will not be used for other studies without the explicit permission of the participant and the approval of the CEIC.

#### 12.4 Insurance

There will be civil liability insurance policy for the trial as established in article 8 of RD 1090/2015, of December 4.

#### 13 PRACTICAL CONSIDERATIONS

#### 13.1 Responsibilities of participants in the study

#### Rules for participants

Participating subjects must follow the indications of the investigators and communicate any eventuality to them.

Participants will be duly informed of the prohibitions or restrictions to which they must be adherent throughout the study. Failure to comply with these recommendations will imply abandoning the study.

All subjects participating in the study have the right to leave the study at any time, withdrawing their consent, without having to justify this decision and without causing any detriment effect in their clinical follow-up. If this occurs, the investigator will try to ensure that the subject performs all the necessary evaluations to ensure that no adverse events occur and to ensure appropriate follow-up.

#### Rules for investigators

Investigators are obliged to comply with the norms established in the current legislation regarding clinical trials.

#### Protocol compliance

Protocol deviations should be avoided. If these occur, the investigator must inform the



monitor and the implications of such deviations will be reviewed and discussed among the investigation team. Deviations from the protocol will be documented specifying the reasons, date, action taken, and the impact on the participant and the trial. Documentation regarding deviations from the protocol will be stored in the Investigator's Archive.

#### 13.2 Monitoring, auditing and inspection

The study will be monitored by a monitor of SEIMC-GESIDA Foundation, who will prepare an appropriate monitoring plan for the study. Regular visits and phone calls will be made to investigators. During visits, the monitor should review participant and study drug records and documents, and the preservation of said documents. In addition, the monitor should evaluate the study procedures and discuss any problems with the investigator. During the course of the study, audit visits may be carried out in the participating centres. The investigators will allow direct access to the source data / documents for monitoring, auditing or review by the La Paz Research Ethics Commitee (Comité Ético de Investigación Clínica, CEIC) and inspection by the Health Authorities.

#### 13.3 Study documentation

All documentation related to the study (protocol, CRD, informed consent, authorizations...) will be archived during the study in a safe place and easily accessible by the research team. All information contained in clinical, histological, biochemical and molecular reports, observations or other activities are necessary for the reconstruction and evaluation of the study. Examples of these documents are hospital records, laboratory notes, memorandums, participant diary, evaluation checklists, medication dispensing record or other pharmacy documents, recording of data obtained from automated devices, digitized photo files, X-rays, etc.

#### 13.4 Data management

Processing, communication and transfer of personal data of all participating subjects will comply with the provisions of Organic Law 03/2018, on the protection of personal data. At the time of registration, a Participant Number will be assigned to each participant. This information will be registered in the CRD. The investigator will be responsible for keeping the appropriate information about each participant so that health authorities can have



access to such information if necessary. These records must be kept confidential for the period of time legally mandated by current regulations.

#### 13.5 Publication conditions

All information from the study will be considered confidential. The Principal Investigator assumes the set of responsibilities linked to this function, and the exclusive ownership of the results of the study, which may be freely exploited. Principal Investigator commits to publish the results of the study in a scientific journal or to make them available to the public as established by the Declaration of Helsinki, item 36: "Researchers, authors, sponsors, editors and publishers all have ethical obligations with regard to the publication and dissemination of the results of research. Researchers have a duty to make publicly available the results of their research on human subjects and are accountable for the completeness and accuracy of their reports. All parties should adhere to accepted guidelines for ethical reporting. Negative and inconclusive as well as positive results must be published or otherwise made publicly available. Sources of funding, institutional affiliations and conflicts of interest must be declared in the publication. Reports of research not in accordance with the principles of this Declaration should not be accepted for publication".

#### 13.6 Procedure for the modifications of the protocol

Any protocol modifications must be documented with a protocol amendment. Amendments will be duly identified by their chronological order number, dated and signed by the sponsor and the investigator. If the modifications are relevant, the sponsor must request authorization from the Reference CEIC and the AEMPS, as established by current regulations.

#### 13.7 Ethics committee of research with medicines (CEIC)

The protocol and the informed consent documents will be evaluated by the CEIC of La Paz University Hospital whose composition is already known and accredited by the health authorities of the Autonomous Community of Madrid (http://www.msssi.gob.es/profesionales/ pharmacy / ceic / pdf / ceicsacreditadoses.pdf). The decision of the CEIC regarding the development of the study will be provided in writing to the investigator. A copy of that decision must be sent to the sponsor.



The sponsor will present the required progress reports of the study to the CEIC and will communicate the suspicions of serious and unexpected adverse reactions. Upon completion of the study, the sponsor must inform the CEIC.

#### 14 STATISTICAL ANALYSIS

#### 14.1 Sample size estimation

In previous studies of switch to DTG/3TC the rate of virologic failure at week 48 has been 0.7%<sup>24</sup>. With 120 participants recruited, and considering the same proportion of virologic failures, we could discard differences in the proportion of virologic failures >4% with a binomial estimation of the 95 confidence interval.

#### 14.2 Statistical analysis

In addition to main analysis, a security analysis will take place at week 24, to determine if study is to be continued (section 7.5).

To compare two means we will use Student's t test (if normal distribution) or non-parametric Wilcoxon rank-sum (Mann-Whitney) test. If needed, an adjusted analysis would be performed. Proportions will be compared with x2 test.

Endpoints will be analysed including the intention-to-treat exposed population, that is, all participants who received at least one dose study drug.

#### Main Analysis – Primary endpoint:

The main primary endpoint will be the proportion of virological failure HIV-1 RNA VL≥50 copies/mL, at 48 weeks, following FDA snapshot algorithm in the population "by intention to treat -exposed". This result will be expressed as a percentage and 95% confidence interval.

#### Secondary planned analysis -Secondary endpoints:

- a. Proportion of VF (≥50 copies/mL) at week 96, ITT-e, FDA snapshot. This result will be expressed as a percentage and 95% confidence interval.
- b. Proportion of VF (≥50 copies/mL) at week 48 and 96, PP population, FDA snapshot.
- c. Proportion of VF (≥200 copies/mL) at week 48 and 96, ITT-e and PP population, FDA snapshot. This result will be expressed as a percentage and 95% confidence interval.



- d. Proportion of CVW at weeks 48 and 96, ITT-e and PP population, FDA snapshot. This result will be expressed as a percentage and 95% confidence interval.
- e. Proportion of PVW at weeks 48 and 96 ITT-e and PP population, FDA snapshot. This result will be expressed as a percentage and 95% confidence interval.
- f. Proportion of participants with VL<50 copies/mL week 48 and 96, ITT-e and PP population, FDA snapshot. This result will be expressed as a percentage and 95% confidence interval.
- g. Incidence of VF with drug resistance associated mutations. Descriptive analysis of number and type of resistance mutations.
- h. Univariant and multivariant logistic regression analysis of factors associated to virological failure (time to VF).
- i. Proportion of VF in pre-specified subgroups:
  - Confirmed historical M184V/I vs No resistance mutations.
  - INSTI exposure vs No prior INSTI exposure.
  - Time virologically suppressed.
  - Time on 3TC/FTC.
- j. Proportion of participants with VF with baseline 3TC or INSTI resistance- associated mutations detected at baseline by NGS with 1, 5, and 20% threshold.
- k. Proportion of participants with transient viral rebounds with baseline 3TC or INSTI resistance- associated mutations detected at baseline by NGS with 1, 5, and 20% threshold.
- Univariant and multivariant logistic regression model analysis of the association between 3TC or integrase resistance-associated mutations by NGS and potentially confounding variables reaching signification below 0.1 in the different univariant models.
- m. Logistic regression model analysis of the impact in virological response of mutations detected by NGS.
- Type and frequency of resistance mutations (RT and integrase) in proviral DNA by NGS at baseline and week 96. Hypermutation analysis of mutations detected through NGS.
- o. Univariant and multivariant logistic regression analysis of factors associated to change on frequency of resistance mutations detected by NGS at baseline and week 96.



- p. Incidence and severity of AEs and laboratory abnormalities grade III-IV through week 48 and 96.
- q. Proportion of subjects who discontinue treatment due to AEs through weeks 48 and 96.
- r. Change from Baseline in CD4<sup>+</sup> cell count (W48 minus baseline and W96 minus W48) and in CD4<sup>+</sup>/CD8<sup>+</sup> cell counts ratio at weeks 48 and 96.

#### 15. REFERENCES

- 1. EACS Guidelines version 10.1, October 2020. 2020. doi:10.1111/fcre.12520
- van Wyk J, Ajana F, Bisshop F, et al. Efficacy and Safety of Switching to Dolutegravir/Lamivudine Fixed-Dose Two-Drug Regimen Versus Continuing a Tenofovir Alafenamide—Based Three- or Four-Drug Regimen for Maintenance of Virologic Suppression in Adults With HIV-1: Phase 3, Randomized, Non-inf. Clin Infect Dis. 2020;53(9):1-30. doi:10.1093/cid/ciz1243
- Charpentier C, Montes B, Perrier M, Meftah N, Reynes J. HIV-1 DNA ultra-deep sequencing analysis at initiation of the dual therapy dolutegravir lamivudine in the maintenance DOLULAM pilot study. *J Antimicrob Chemother*. 2017;72(10):2831-2836. doi:10.1093/jac/dkx233
- Baldin G, Ciccullo A, Borghetti A, Di Giambenedetto S. Virological efficacy of dual therapy with lamivudine and dolutegravir in HIV-1-infected virologically suppressed patients: long-term data from clinical practice. *J Antimicrob* Chemother. 2019;74(5):1461-1463. doi:10.1093/jac/dkz009
- Gagliardini R, Ciccullo A, Borghetti A, et al. Impact of the M184V Resistance Mutation on Virological Efficacy and Durability of Lamivudine-Based Dual Antiretroviral Regimens as Maintenance Therapy in Individuals With Suppressed HIV-1 RNA: A Cohort Study. Open Forum Infect Dis. 2018;5(6):1-8. doi:10.1093/ofid/ofy113
- 6. De Miguel R, Rial-Crestelo D, Dominguez-Dominguez L, et al. Dolutegravir plus lamivudine for maintenance of HIV viral suppression in adults with and without historical resistance to lamivudine: 48-week results of a non-randomized, pilot clinical trial (ART-PRO). *EBioMedicine*. 2020;55:102779. doi:10.1016/j.ebiom.2020.102779



- Rial-Crestelo D, de Miguel R, Montejano R, et al. Long-term efficacy of dolutegravir plus lamivudine for maintenance of HIV viral suppression in adults with and without historical resistance to lamivudine: Week 96 results of ART-PRO pilot study. *J Antimicrob Chemother*. November 2020:1-5. doi:10.1093/jac/dkaa479
- 8. EACS Guidelines version 10.0, November 2019. 2019; (November).
- 9. Cahn P, Madero JS, Arribas JR, et al. Dolutegravir plus lamivudine versus dolutegravir plus tenofovir disoproxil fumarate and emtricitabine in antiretroviral-naive adults with HIV-1 infection (GEMINI-1 and GEMINI-2): week 48 results from two multicentre, double-blind, randomised, non-inferior. *Lancet*. 2019;393(10167):143-155. doi:10.1016/S0140-6736(18)32462-0
- 10. World Health Organization (WHO). *HIV Drug Resistance Report*.; 2019. http://scholar.google.com/scholar?hl=en&btnG=Search&q=intitle:Who+hiv+drug +resistance+report+2012#5.
- 11. Ciaffi L, Koulla-Shiro S, Sawadogo AB, et al. Boosted protease inhibitor monotherapy versus boosted protease inhibitor plus lamivudine dual therapy as second-line maintenance treatment for HIV-1-infected patients in sub-Saharan Africa (ANRS12 286/MOBIDIP): a multicentre, randomised, parallel, open-la. Lancet HIV. 2017;4(9):e384-e392. doi:10.1016/S2352-3018(17)30069-3
- Gregson J, Tang M, Ndembi N, et al. Global epidemiology of drug resistance after failure of WHO recommended first-line regimens for adult HIV-1 infection: a multicentre retrospective cohort study. *Lancet Infect Dis.* 2016;16(5):565-575. doi:10.1016/S1473-3099(15)00536-8
- Pouga L, Santoro MM, Charpentier C, et al. New resistance mutations to nucleoside reverse transcriptase inhibitors at codon 184 of HIV-1 reverse transcriptase (M184L and M184T). Chem Biol Drug Des. 2019;93(1):50-59. doi:10.1111/cbdd.13378
- Domínguez-Domínguez L, Montejano R, Esteban-cantos A, et al. Prevalence and factors associated to the detection (population and next generation sequencing) of archived 3TC resistance mutations in aviremic HIV-infected adults (GEN-PRO). GeSIDA. 2019;3(3):837.
- 15. Wirden M, Soulie C, Valantin MA, et al. Historical HIV-RNA resistance test results are more informative than proviral DNA genotyping in cases of suppressed or

VOLVER Study protocol 4.0, 31 May 2021



- residual viraemia. *J Antimicrob Chemother*. 2011;66(4):709-712. doi:10.1093/jac/dkq544
- Allavena C, Rodallec A, Leplat A, et al. Interest of proviral HIV-1 DNA genotypic resistance testing in virologically suppressed patients candidate for maintenance therapy. J Virol Methods. 2018;251(October 2017):106-110. doi:10.1016/j.jviromet.2017.10.016
- Delaugerre C, Braun J, Charreau I, et al. Comparison of resistance mutation patterns in historical plasma HIV RNA genotypes with those in current proviral HIV DNA genotypes among extensively treated patients with suppressed replication. HIV Med. 2012;13(9):517-525. doi:10.1111/j.1468-1293.2012.01002.x
- Dauwe K, Staelens D, Vancoillie L, Mortier V, Verhofstede C. Deep Sequencing of HIV-1 RNA and DNA in Newly Diagnosed Patients with Baseline Drug Resistance Showed No Indications for Hidden Resistance and Is Biased by Strong Interference of Hypermutation. Caliendo AM, ed. *J Clin Microbiol*. 2016;54(6):1605-1615. doi:10.1128/JCM.00030-16
- Ho YC, Shan L, Hosmane NN, et al. Replication-competent noninduced proviruses in the latent reservoir increase barrier to HIV-1 cure. Cell. 2013;155(3):540. doi:10.1016/j.cell.2013.09.020
- 20. Paton NI, Kityo C, Hoppe A, et al. Assessment of second-line antiretroviral regimens for HIV therapy in Africa. *N Engl J Med.* 2014;371(3):234-247. doi:10.1056/NEJMoa1311274
- La Rosa AM, Harrison LJ, Taiwo B, et al. Raltegravir in second-line antiretroviral therapy in resource-limited settings (SELECT): a randomised, phase 3, noninferiority study. *Lancet HIV*. 2016;3(6):e247-e258. doi:10.1016/S2352-3018(16)30011-X
- 22. SECOND LINE Study Group. Ritonavir-boosted lopinavir plus nucleoside or nucleotide reverse transcriptase inhibitors versus ritonavir-boosted lopinavir plus raltegravir for treatment of HIV-1 infection in adults with virological failure of a standard first-line ART regimen (SECOND. *Lancet*. 2013;381(9883):2091-2099. doi:10.1016/S0140-6736(13)61164-2
- 23. Wyk J Van, Ajana F, Bisshop F, et al. Switching To DTG-3TC Fixed-Dose Combination (Fdc) Is Non-Inferior To Continuing a Taf-Based Regimen in Maintaining Virologic Suppression Through 48 Weeks (Tango Study). IAS 2019.



2019.

- 24. Wandeler G, Buzzi M, Anderegg N, et al. Virologic failure and HIV drug resistance on simplified, dolutegravir-based maintenance therapy: Systematic review and meta-analysis. F1000Research. 2018;7(0):1359. doi:10.12688/f1000research.15995.2
- 25. World Medical Association. Declaration of Helsinki- Ethical principles for medical research involving human subjects. *World Med Assoc.* 2013.
- 26. Perrier M, Visseaux B, Landman R, et al. No impact of HIV-1 protease minority resistant variants on the virological response to a first-line PI-based regimen containing darunavir or atazanavir. *J Antimicrob Chemother*. 2018;73(1):173-176. doi:10.1093/jac/dkx366
- 27. Schmieder R, Edwards R. Quality control and preprocessing of metagenomic datasets. *Bioinformatics*. 2011;27(6):863-864. doi:10.1093/bioinformatics/btr026
- 28. Magoč T, Salzberg SL. FLASH: Fast length adjustment of short reads to improve genome assemblies. *Bioinformatics*. 2011;27(21):2957-2963. doi:10.1093/bioinformatics/btr507
- 29. De Miguel Buckley R, Rial-Crestelo D, Dominguez-Dominguez L, et al. Dolutegravir ( DTG ) and Lamivudine ( 3TC ) for Maintenance of HIV Viral Suppression in Adults With and Without Historical Resistance to Lamivudine: 48- Week Results of a Pilot Clinical Trial (ART-PRO). In: European AIDS Conference.
- Dovato. Summary of product characteristics. Eur Med Agency. 2019. doi:10.2307/j.ctvdf0dxq.12
- 31. U.S. Department of Health and Human Services, National Institutes of Health, National Institute of Allergy and Infectious Diseases Division of AIDS. Division of AIDS (DAIDS) Table for Grading the Severity of Adult and Pediatric Adverse Events, Corrected Version 2.1. [July 2017]. Natl Inst Allergy Infect Dis. 2017. https://rsc.niaid.nih.gov/sites/default/files/daidsgradingcorrectedv21.pdf.



#### APPENDIX 1. GUIDANCE ON PREGNANCY AND BREAST FEEDING

Preliminary results from an observational study revealed an increased risk of neural tube defects in infants born to women who took dolutegravir at the time of conception. Later data from the study has shown a numerically higher rate of neural tube defects with exposure to dolutegravir compared to non-dolutegravir-containing antiretroviral regimens at the time of conception, however, the difference was not statistically significant. A causal relationship of these events to the use of dolutegravir has not been established. No increased risk was reported in infants born to women who started dolutegravir later during pregnancy.

Reproductive toxicology studies have not shown any relevant findings. Likewise, other data on the use of dolutegravir in pregnancy, including data from the Antiretroviral Pregnancy Registry (APR), clinical trials and post-marketing use have not indicated an increased risk of neural tube defects, although the extent of exposure from these other data sources is currently insufficient to confirm or rule out an increased risk of neural tube defects with DTG-containing regimens taken at the time of conception and in early pregnancy.

Further information about this potential risk is provided in the Investigator Brochure for DTG-containing products and, where applicable, the approved Local Prescribing Information).

Reproductive toxicity data for 3TC and DTG guidance on the use of these active principle in pregnancy, is given in the relevant approved Local Prescribing Information.

A female, may be eligible to enter and participate in the study if she:

- a. is of non-child-bearing potential defined as either post-menopausal (12 months of spontaneous amenorrhea and ≥45 years of age) or physically incapable of becoming pregnant with documented tubal ligation, hysterectomy or bilateral oophorectomy or,
- is of child-bearing potential with a negative pregnancy test at both Screening and Visit 1 and agrees to use one of the highly effective methods to avoid pregnancy documented below.



Women of childbearing potential should be informed about the potential risk of neural tube disorders with DTG. These defects happen early in pregnancy, before many women even know they are pregnant.

Women of childbearing potential should be counselled about the importance of pregnancy avoidance, safer sexual practices and adherence to contraception requirements throughout the study, and for at least 4 weeks after the last study visit.

Women of childbearing potential must be using a highly effective method of contraception as detailed below, which should be documented in the eCRF.

Females of childbearing potential should be reminded about the importance of pregnancy avoidance and of adherence to contraception requirements at every study visit.

If pregnancy is confirmed while taking DTG/3TC, treatment should be discontinued and the subject should be switched to an alternative regimen

Highly Effective Methods for Avoiding Pregnancy in Females of Reproductive potential:

- Complete abstinence from penile-vaginal intercourse from 2 weeks prior to administration
  of Investigational Product, throughout the study, and for at least 4 weeks after
  discontinuation of all study medications;
- Any intrauterine device with published data showing that the expected failure rate is <1% per year:

Implantable progestogen-only hormonal contraception associated with inhibition of ovulation

Intrauterine device (IUD)

Intrauterine hormone-releasing system (IUS)

bilateral tubal occlusion.

- Male partner sterilization confirmed prior to the female subject's entry into the study, and this male is the sole partner for that subject;
- Approved hormonal contraception:

Combined (estrogen- and progestogen-containing) hormonal contraception associated with inhibition of ovulation: oral intravaginal or transdermal.



to Sponsor.



Progestogen-only hormonal contraception associated with inhibition of ovulation: injectable.

Any other method with published data showing that the expected failure rate is <1% per year.</li>

Any contraception method must be used consistently, in accordance with the approved product label and for at least 4 weeks after discontinuation of study medication.

#### Reporting of pregnancy information

Any pregnancy that occurs during study participation must be reported (see Appendix 5 and 6). To ensure subject safety, each pregnancy must be reported to Sponsor within 24 hours of learning of its occurrence. All pregnancies should also be reported to ViiV Healthcare within 1 week, regardless of causality. The pregnancy must be followed up to determine outcome (including premature termination) and status of mother and child, which must also be reported to Sponsor. Pregnancy complications and elective terminations for medical reasons must be reported as an adverse event or serious adverse event. Spontaneous abortions must be reported as a serious adverse event. Any serious adverse event occurring in association with a pregnancy brought to the investigator's attention after the subject has completed the study and considered by the

Investigators are also encouraged to report any pregnancy that occurs during study participation to the Antiretroviral Pregnancy Registry (APR) prospectively, and before the pregnancy outcome. More information including copies of applicable case report forms and fax numbers are available at www.apregistry.com.

investigator as possibly related to the investigational product, must be promptly reported



#### APPENDIX 2: RISK ASSESSMENT AND TOXICITY MANAGEMENT

Reference safety information for this study is the Investigator Brochure and/or approved Local Prescribing Information for the study treatments.

Here we summarized some risk and toxicity information, especially of DTG.

The current key risks associated with the use of the DTG single entity or other DTG-containing products are presented below. Further information on these, and other known or theoretical risks associated with the use of these products, is included in the Investigator Brochure for the DTG-containing products, and, where applicable, in the approved Local Prescribing Information.

#### Risk Assessment

| Potential Risk of<br>Clinical<br>Significance | Data/Rationale for Risk | Mitigation Strategy |
|---|---|---|
| Refer to Invest | Investigational Product: dolutegravi<br>igator Brochure and/or approved Loca<br>additional information | |
| Hypersensitivity and rash | Hypersensitivity reactions has been observed uncommonly with DTG. Rash, generally mild to moderate in intensity, was commonly reported in DTG Phase IIb/III clinical trials. No episodes of severe rash, such as Stevens-Johnson Syndrome, toxic epidermal necrolysis and erythema multiforme, were reported. | Subjects with history or presence of allergy to any of the study drugs or their components are excluded. Specific/detailed toxicity management guidance is provided for hypersensitivity reactions and rash. The subject informed consent form includes information on this risk and the actions subjects should take in the event of a hypersensitivity reaction or associated signs and symptoms. |



| GESIDA 11820 | | FUNDACION<br>SEIMC-GESIDA |
|---|---|---|
| Potential Risk of<br>Clinical<br>Significance | Data/Rationale for Risk | Mitigation Strategy |
| Refer to Investi | Investigational Product: dolutegravi<br>gator Brochure and/or approved Loca<br>additional information | |
| Drug induced liver injury and | Non-clinical data suggested a possible, albeit low, risk for | Subjects meeting any of the following criteria during the |
| other clinically significant liver chemistry elevations | possible, albeit low, risk for hepatobiliary toxicity with DTG. Drugrelated hepatitis is considered an uncommon risk for antiretroviral therapy containing DTG regardless of dose or treatment population. For subjects with hepatitis B virus and/or hepatitis C virus co-infection, improvements in immunosuppression because of human immunodeficiency virus (HIV) virologic and immunologic responses to DTG-containing antiretroviral therapy, along with inadequate therapy for hepatitis B virus co-infected subjects, likely contributed to significant elevations in liver chemistries. There have been rare post-marketing reports of acute hepatic failure in association with DTG-containing regimens. Current treatment guidelines do not recommend mono-therapy with 3TC for patients with hepatitis B virus infection, which is what subjects on | following criteria during the screening period are excluded from participating • Alanine aminotransferase (ALT) ≥ 5 times the upper limit of normal (ULN) or ALT ≥ 3xULN and bilirubin ≥1.5xULN (with >35% direct bilirubin) • Unstable liver disease, cirrhosis and/or known biliary abnormalities (except for hyperbilirubinemia or jaundice due to Gilbert's syndrome or asymptomatic gallstones) • Subjects with an anticipated need for hepatitis C virus therapy with interferon and/or ribavirin prior to the primary endpoint • Positive Surface Hepatitis B Ag (HBAgS) OR negative HBAgS and negative hepatitis B surface antibody (anti-HBs) with positive anticore antibody (anti-HBc) and positive HBV DNA. • Specific/detailed liver stopping criteria and toxicity management guidance is provided for suspected drug induced liver injury or other clinically significant liver chemistry elevations |

Emergence

of HBV

variants



| Potential Risk of<br>Clinical<br>Significance | Data/Rationale for Risk | Mitigation Strategy |
|---|---|---|
| Refer to Invest | Investigational Product: dolutegravi<br>igator Brochure and/or approved Loca<br>additional information | |
| | associated with resistance to 3TC has been reported in HIV-1-infected patients who have received 3TC-containing antiretroviral regimens in the presence of concurrent infection with HBV. Additionally, discontinuation of 3TC in hepatitis B virus infected subjects can result in severe exacerbations of hepatitis B virus. For subjects co-infected with hepatitis C virus and HIV, [some] treatment guidelines recommend that the hepatitis C virus infection is treated first before starting treatment for the HIV. Additionally, interferon and/or ribavirin toxicity maybe frequent and difficult to differentiate causality from investigational product. | |
| Theoretical serious drug interaction with dofetilide and pilsicainide | Dolutegravir must not be administered concurrently with medicinal products with narrow therapeutic windows, that are substrates of organic cation transporter 2 (OCT2), including but not limited to dofetilide, pilsicainide or fampridine (also known as dalfampridine. | The co-administration of DTG/3TC with dofetilide or fampridine are prohibited in the study. |
| Psychiatric disorders | Psychiatric disorders including suicide ideation and behaviours are | Due to the elevated risk in the HIV-infected population, |



| Potential Risk of<br>Clinical<br>Significance | Data/Rationale for Risk | Mitigation Strategy |
|---|---|---|
| Refer to Investi | Investigational Product: dolutegravir/lamivudine Refer to Investigator Brochure and/or approved Local Prescribing Information for additional information | |
| | common in HIV-infected patients. In clinical trials, the psychiatric profile for DTG (including suicidality, depression, bipolar and hypomania, anxiety and abnormal dreams) was generally similar or favourable compared with other antiretroviral therapy, although a higher incidence of depression and suicidal ideation /behaviours with DTG compared with darunavir/ritonavir was noted in the FLAMINGO clinical study. An evaluation of aggregate data, including post-marketing data concluded that a causal association between DTG and depression and suicidal behaviours could not be ruled out. These events occur primarily in patients with a prior history of psychiatric illness. The reporting rate for insomnia was statistically higher for blinded DTG+ABC/3TC compared to efavirenz/tenofovir/emtricitabine in the SINGLE clinical study; however, this was not duplicated in other VH Sponsored Phase IIb/III studies with | treatment emergent assessment of suicidality will be monitored during this study. Investigators are advised to consider mental health consultation or referral for subjects who experience signs of suicidal ideation or behaviour |



| Potential Risk of<br>Clinical<br>Significance | Data/Rationale for Risk | Mitigation Strategy |
|---|---|---|
| | Investigational Product: dolutegravir/lamivudine<br>Refer to Investigator Brochure and/or approved Local Prescribing Information for<br>additional information | |
| Renal function | Lamivudine is eliminated by renal excretion and exposure increases in patients with renal dysfunction. | Due to requirements for dose reduction of 3TC in patients with renal dysfunction, subjects with a creatinine clearance <30 mL/min (CKD-EPI method) are excluded. Participants who develop a Grade 4 eGFR toxicity (per DAIDs criteria) should have study drug withdrawn. |
| Neural tube defects | In a birth surveillance study conducted in Botswana (the Tsepamo study), preliminary results showed that in babies born to women who were taking DTG when they became pregnant there was an increased risk of neural tube defects compared with the background rate. Later data from the study has shown a numerically higher rate of neural tube defects with exposure to DTG compared to non-DTG-containing antiretroviral regimens at the time of conception, however, the difference was not statistically significant. A causal relationship of these events to the use of DTG has not been established. No increased risk of these defects was reported in babies born to mothers | Pregnancy testing should be performed before initiation of DTG therapy in all women of childbearing potential (negative pregnancy test at screening and randomization). (Section 9) Women who are pregnant or who plan to become pregnant, are excluded. All women of reproductive potential should use a highly effective method of contraception – see Section11.7 /Appendix 1 Subject informed consent form provides information about this potential risk. |



| Potential Risk of<br>Clinical<br>Significance | Data/Rationale for Risk | Mitigation Strategy |
|---|---|---|
| Investigational Product: dolutegravir/lamivudine<br>Refer to Investigator Brochure and/or approved Local Prescribing Information for<br>additional information | | |
| | who started DTG containing regimen | |
| | later in pregnancy | |
| | Dolutegravir was tested in a complete package of reproductive toxicology studies, including embryofoetal development studies. No adverse development outcomes, including neural tube defects, were identified. In reproductive toxicity studies in animals, DTG was shown to cross the placenta. Data analysed to date from other sources including the Antiretroviral Pregnancy Registry, clinical trials, and post-marketing data are insufficient to address the risk of neural tube defects with DTG. | |

#### **Toxicity Management**

In the event of a discontinuation of a DTG-containing product for suspected drug induced liver injury, other clinically significant liver chemistry elevations, severe skin reaction or hypersensitivity reaction, subjects should not be rechallenged with a DTG-containing product due to the risk of a recurrent reaction. These subjects should be withdrawn from study and seek/be reviewed for alternative antiretroviral therapy (but may continue on study, but off study drug). Further details on this are provided in this section as appropriate.

#### Hypersensitivity and rash





#### Allergic Reaction

Subjects may continue investigational product(s) for Grade 1 or 2 allergic reactions at the discretion of the Investigator. The subject should be advised to contact the Investigator immediately if there is any worsening of symptoms or if further systemic signs or symptoms develop. Antihistamines, topical corticosteroids, or antipruritic agents may be prescribed.

Subjects with Grade ≥3 allergic reactions that are considered to be possibly or probably related to the investigational product(s) should permanently discontinue the investigational product regimen and the subject should be withdrawn from the study. Subjects should be treated as clinically appropriate and followed until resolution of the adverse event.

#### Rash

Mild to moderate rash is an expected adverse reaction for DTG-containing antiretroviral therapy. Episodes generally occur within the first ten weeks of treatment, rarely require interruptions or discontinuations of therapy and tend to resolve within two to three weeks. The index case of a hypersensitivity reaction with DTG involved a profuse, purpuric and coalescing leukocytoclastic vasculitis as well as clinically significant liver chemistry elevations. Other than this case, no other instances of serious skin reaction, including Stevens-Johnson Syndrome, toxic epidermal necrolysis and erythema multiforme have been reported for DTG in clinical trials.

Subjects with an isolated Grade 1 rash may continue investigational product at the Investigator's discretion. The subject should be advised to contact the Investigator immediately if there is any worsening of the rash, if any systemic signs or symptoms worsen, or if mucosal involvement develops.

Subjects may continue investigational product for an isolated Grade 2 rash. However, investigational product (and all other concurrent medication(s) suspected in the Investigators causality assessment) should be permanently discontinued for any Grade ≥2 rash that is associated with an increase in ALT. The subject should be advised to contact the physician immediately if rash fails to resolve (after more than two weeks), if there is any worsening of the rash, if any systemic signs or allergic symptoms develop, or if mucosal involvement develops.



Subjects should permanently discontinue investigational product (and all other concurrent medication(s) suspected in the Investigators causality assessment) for an isolated Grade 3 or 4 rash, and the subject should be withdrawn from the study. Subjects should be treated as clinically appropriate and followed until resolution of the adverse event.

The rash and any associated symptoms should be reported as adverse events (see (Section 11) and appropriate toxicity ratings should be used to grade the events (based on DAIDS [Division of ADS] toxicity gradings).

If the etiology of the rash can be diagnosed as being unrelated to investigational product and due to a specific medical event or a concomitant non-study medication, routine management should be performed and documentation of the diagnosis provided.

#### • Liver Chemistry Stopping and Follow up Criteria

Liver chemistry stopping and increased monitoring criteria have been designed to assure subject safety and evaluate liver event etiology during administration of study drug and the follow-up period (in alignment with the FDA premarketing clinical liver safety quidance).

http://www.fda.gov/downloads/Drugs/GuidanceComplianceRegulatoryInformation/Guidances/UCM174090.pdf

For any participant meeting one of the criteria outlined in Table 1 or <u>Table 2</u>, or if the Investigator believes that it is in the best interest of the patients, the Investigator must follow the required actions and follow up assessments also outlined in these tables.

Table 1 Liver Chemistry Stopping Criteria - Liver Stopping Event

| ALT absolute | ALT ≥ 8xULN |
|---|---|
| ALT increase | ALT ≥ 5xULN but <8xULN persists for ≥2 weeks (with bilirubin <2xULN and no signs or symptoms of acute hepatitis or hypersensitivity) |
| Bilirubin <sup>1, 2</sup> | ALT ≥ 3xULN and bilirubin ≥ 2xULN (>35% direct bilirubin) |
| INR <sup>2</sup> | ALT ≥ 3xULN <b>and</b> International normalised ratio (INR)>1.5, if INR measured |
| Cannot<br>Monitor | ALT ≥ 5xULN but <8xULN and cannot be monitored weekly for >2 weeks |



| GESIDA 11820 | | SEIMC-GESIDA • |
|---|---|---|
| | (See Table 2 for actions when weeks) | re subjects CAN be monitored weekly for >2 |
| Symptomatic <sup>3</sup> | ALT ≥ 3xULN (if baseline ALT believed to be related to liver in | is □ULN) with symptoms (new or worsening)<br>njury or hypersensitivity |
| | ALT ≥ 3x baseline (if baseline Abelieved to be related to liver in | ALT>ULN) with symptoms (new or worsening)<br>njury or hypersensitivity |
| Required Ac | tions and Follow up Assessme | ents following ANY Liver Stopping Event |
| | Actions | Follow Up Assessments |
| <ul> <li>Immediately</li> </ul> | / hold DTG. | Viral hepatitis serology, including: |
| event and I | relationship between the liver<br>DTG cannot be ruled out, then | <ul> <li>Hepatitis A immunoglobulin M<br/>(IgM) antibody;</li> </ul> |
| and the Sub | be permanently discontinued<br>iject not rechallenged due to the<br>urrent reaction. | <ul> <li>HBsAg and hepatitis B core<br/>antibody;</li> </ul> |
| | e event to the Sponsor by | Hepatitis C RNA; |
| · | vithin 24 hours. | Hepatitis E IgM antibody. |
| with hyperb<br>Sponsor as<br>the serious | ossible drug-induced liver injury ilirubinemia <sup>2</sup> will be reported to serious adverse events using adverse event case report form. | <ul> <li>Cytomegalovirus IgM antibody.</li> <li>Epstein-Barr viral capsid antigen IgM antibody (or if unavailable, obtain heterophile antibody or monospot</li> </ul> |
| for all event<br>and submit | ne liver event case report form<br>s meeting liver stopping criteria,<br>to Sponsor within one week of<br>ng aware of the event | <ul><li>testing).</li><li>Syphilis screening.</li><li>Drugs of abuse screen, including</li></ul> |
| Perform live | er event follow up assessments. | alcohol. Record alcohol use on the liver event case report form |
| resolve, st | subject until liver chemistries cabilise, or return to within the MONITORING below). | Serum acetaminophen adduct High<br>Performance Liquid Chromatography |
| alternative of<br>liver injury,<br>considered<br>Liver Sat | event has a clear underlying cause, other than drug-induced then Drug Restart may be by Sponsor (for exception see fety – Study Treatment e and Restart) | assay (quantifies potential acetaminophen contribution to liver injury in subjects with definite or likely acetaminophen use in the preceding week (2) [FDA, 2009]). The site must contact the medical monitor when this test is required. NOTE: not required in |
| permanently | · | <ul> <li>China</li> <li>Serum creatinine kinase and lactate dehydrogenase.</li> <li>Fractionate bilirubin, if total bilirubin ≥1.5xULN.</li> </ul> |
| MONITORING: | | Obtain complete blood count with |
| | reasonable attempt to have urn to clinic within 24 hours for | differential to assess eosinophilia. |

subjects return to clinic within 24 hours for repeat liver chemistries (include ALT,



- aspartate aminotransferase, alkaline phosphatase, bilirubin) and perform liver event follow up assessments at the central laboratory as described to the right.
- A specialist or hepatology consultation is recommended.
- Monitor subjects twice weekly until liver chemistries resolve, stabilise or return to within baseline.
- Anti-nuclear antibody, anti-smooth muscle antibody, Type 1 anti-liver kidney microsomal antibodies, and quantitative total immunoglobulin G (or gamma globulins).
- Liver imaging (ultrasound, magnetic resonance, or computerised tomography) and /or liver biopsy to evaluate liver disease. Complete Liver Imaging and/or Liver Biopsy case report form.
- Record use of concomitant medications on the concomitant medications report form including acetaminophen, herbal remedies, other over the counter medications.
- 1. Serum bilirubin fractionation should be performed if testing is available. If serum bilirubin fractionation is not immediately available, discontinue study treatment for that subject if ALT ≥ 3xULN and bilirubin ≥ 2xULN. Additionally, if serum bilirubin fractionation testing is unavailable, record presence of detectable urinary bilirubin on dipstick, indicating direct bilirubin elevations and suggesting liver injury.
- 2. All events of ALT ≥ 3xULN and bilirubin ≥ 2xULN (>35% direct bilirubin) or ALT ≥ 3xULN and INR>1.5, if INR measured which may indicate severe liver injury must be reported as a serious adverse event (excluding studies of hepatic impairment or cirrhosis); INR measurement is not required and the threshold value stated will not apply to subjects receiving anticoagulants
- 3. New or worsening symptoms believed to be related to liver injury (such as fatigue, nausea, vomiting, right upper quadrant pain or tenderness, or jaundice) or believed to be related to hypersensitivity (such as fever, rash or eosinophilia). Record the appearance or worsening of any such clinical symptoms on the adverse event report form.

Table 2 Liver Chemistry Increased Monitoring Criteria

| Criteria | Actions |
|---|---|
| ALT ≥5xULN and <8xULN and bilirubin <2xULN without symptoms believed to be related to liver injury or hypersensitivity, and who can be monitored weekly for >2 weeks. | <ul> <li>Notify the medical monitor within 24 hours of learning of the abnormality to discuss subject safety.</li> <li>Subject can continue study treatment</li> <li>Subject must return weekly for repeat liver chemistries (ALT, aspartate aminotransferase, alkaline phosphatase, bilirubin) until resolution, stabilisation (ALT &lt;5×ULN on 2 consecutive evaluations) or return to within baseline</li> </ul> |



| • | If at any time subject meets the liver chemis | stry |
|---|-----------------------------------------------|------|
| | stopping criteria, proceed as described above | |

#### Liver Safety - Study Treatment Rechallenge and Restart

**Rechallenge** refers to resuming study treatment following drug induced liver injury. Following DILI, drug rechallenge is associated with a 13% mortality across all drugs in prospective studies (1) [Andrade et, 2009]. Clinical outcomes vary by drug, with nearly 50% fatality with halothane readministered within one month of initial injury. However, some drugs seldom result in recurrent liver injury or fatality.

In the event of a discontinuation of DTG/3TC for a Liver Stopping Event, subjects should not be rechallenged with DTG/3TC due to the risks associated with rechallenge.

'Drug restart' refers to resuming study treatment following a Liver Stopping Event in which there is a clear underlying cause (other than drug induced liver injury) of the liver event (e.g. biliary obstruction, pancreatic events, hypotension, acute viral hepatitis). If a causal relationship between the liver event and DTG/3TC cannot be ruled out, then DTG/3TC must be permanently discontinued and the subject not rechallenged. Drug restart with DTG/3TC in a patient who has a Liver Stopping Event is permitted providing the investigator follows the specific Drug Restart Criteria:

## <u>Drug Restart Following Transient Resolving Liver Events Not Related to Study</u> <u>Drug</u>

Restart can be considered when liver chemistries improve to within 1.5x baseline and ALT<3xULN) where:

- Liver chemistries have a clear underlying cause other than drug-induced liver injury (e.g. biliary obstruction, pancreatic events, hypotension, acute viral hepatitis).
   Furthermore, there should be no evidence of alcoholic hepatitis or hypersensitivity, and the drug should not be associated with HLA markers of liver injury.
- The subject is receiving compelling benefit and benefit of drug restart exceeds risk
- Approval from Study Team and Ethics Committee or Institutional Review Board for the drug restart has been obtained.



- The subject has been provided with a clear description of the possible benefits and risks of drug restart, including the possibility of recurrent, more severe liver injury or death.
- The subject has also provided signed informed consent specifically for the restart.
   Documentation of informed consent must be recorded in the study file.
- Following drug restart, the Subject will return to the clinic once a week for liver chemistry tests for one month or for as long as clinically indicated and then laboratory monitoring may resume as per protocol. If protocol defined stopping criteria for liver chemistry elevations are met, study drug must be stopped.

See Appendix 3. Liver safety -Checklist for Drug Restart Approval or Refusal.

#### **Suicidal Risk Monitoring**

Subjects with HIV infection may occasionally present with symptoms of depression and/or suicidality (suicidal ideation or behaviour). In addition, there have been some reports of depression, suicidal ideation and behaviour (particularly in patients with a pre-existing history of depression or psychiatric illness) in some patients being treated with integrase inhibitors, including DTG. Therefore, it is appropriate to monitor subjects for suicidality before and during treatment.

Subjects should be monitored appropriately and observed closely for suicidal ideation and behaviour, or any other unusual changes in behaviour. It is recommended that the investigator consider mental health consultation or referral for subjects who experience signs of suicidal ideation or behaviour.

If any subject experiences a possible suicidality-related adverse event (PSRAE) while participating in this study that is considered by the Investigator to meet ICH E2A (ICH E2A, 1994) definitions for seriousness, the Investigator will collect information using a PSRAE case report form (or agreed alternative) in addition to reporting the event on a serious adverse event case report form. A PSRAE may include, but is not limited to, an event that involves suicidal ideation, a preparatory act toward imminent suicidal behaviour, a suicide attempt, or a completed suicide. The investigator will exercise his or her medical and scientific judgment in deciding whether an event is possibly suicide-



related. PSRAE forms should be completed and reported to Sponsor within one week of the investigator diagnosing a possible suicidality-related serious adverse event.

#### **Decline in Renal Function**

Treatment with DTG/3TC must be discontinued in any Subject developing a grade 4 decreased in creatinine clearance.

A confirmatory creatinine clearance assessment should be conducted within 2 weeks.

#### References:

- 1. Andrade RJ, Robles M, Lucena MI. Rechallenge in drug-induced liver injury: the attractive hazard. Expert Opin Drug Saf. 2009;8:709-714.
- 2. FDA Guidance for Industry Drug-Induced Liver Injury: Premarketing Clinical Evaluation. July 2009. Accessed 07 January 2015 at: http://www.accessdata.fda.gov/drugsatfda\_docs/label/2014/022145s032,203045s010,2 05786s001lbl.pdf
- 3. International Conference on Harmonization of Technical Requirements for Registration of Pharmaceuticals For Human Use. ICH Harmonized Tripartite Guideline. Clinical safety data management: Definitions and standards for expedited reporting. ICH E2A. 1994



#### **APPENDIX 3: Liver Safety – Checklist for Drug Restart Approval or Refusal**

"Drug restart" after discontinuation of Study Drug due to Liver Stopping Criteria (as defined in the protocol), can only be approved by the Study's Governing Body (e.g., Protocol/Study Team or Study Chair) or Principal Investigator for **transient**, **defined non-drug-induced liver injury with no evidence of:** 

- immunoallergic injury/HLA association with injury
- drug-induced liver injury
- · alcoholic hepatitis

#### **Investigators MUST:**

- Hold study drug while labs and evaluations are completed to assess diagnosis, and not restart until "Drug restart" has been approved by the Study's Governing Body or Principal Investigator.
- 2. Complete the table below and submit to the Study's Governing Body or Principal Investigator. The Liver Event case report form should already have been submitted to the Study's Governing Body or Principal Investigator, along with liver imaging and/or liver biopsy case report forms and/or SAE case report form where applicable. Where restart of TRIUMEQ or any other ABC-containing product is being considered, provide documentation verifying HLA-B\*5701 status.

| Subject Number: | Yes | No |
|---|---|---|
| Have liver chemistries improved to within 1.5x baseline and ALT<3xULN? | | |
| Was subject's HIV infection stable or improving on Study Drug? | | |
| Were any of the <b>following high risk factors</b> included in the initial liver injury every <b>(Do not restart if 'Yes' for any one of the following high risk factors)</b> : | ent? | |
| fever, rash, eosinophilia, or hypersensitivity | | |
| drug-induced liver injury | | |
| alcoholic hepatitis (aspartate aminotransferase>ALT, typically <10xULN) | | |
| <ul> <li>Study Drug (other than ABC) has an HLA genetic marker associated with<br/>liver injury</li> </ul> | | |
| For restart of TRIUMEQ, or any other abacavir- containing Study Drug, the subject MUST be HLA-B*5701 negative <sup>1</sup> Specify HLA-B*5701 status <sup>2</sup> : | | |

- In countries/regions where HLA-B\*5701 pre-therapy screening is not considered standard of care, subjects stopping abacavir- containing study drug due to Liver Stopping Criteria MUST be tested and found to be negative for the HLA-B\*5701 allele before abacavir- containing Study Drug can be re-started.
- 2. If study drug does not containing ABC then record HLA-B\*5701 status as "not applicable"



#### **APPENDIX 4: SERIOUS ADVERSE EVENT REPORT FORM**

### SERIOUS ADVERSE EVENT REPORT FORM SEIMC-GESIDA Foundation

| Principal Investigator:<br>Site:<br>Phone: | | | | PROTOCOL CODE (sponsor) EUDRACT N°/ Protocol N° AEMPS | | | □ Initial Report □ Follow up Report | |
|---|---|---|---|---|---|---|---|---|
| Country: NOTIFICATION N° (to be completed by sponsor): | | | | | | | | |
| NOTIFIC. | ATION N° (to | be comp | leted by sp | onsor): | | | | |
| I. INFORM | IATION AB | OUT TH | E ADVER | SE EVENT | W-1" | | 100 | |
| PATIENT<br>CODE: | DATE OF BIRTH AGE (Years): | | □ MALE □ FEMALE | WEIGHT<br>(Kg): | HEIGHT<br>(cm): | SAE START DAT!<br>(dd/mm/yyyy): | SAE START<br>TIME (hh:mm) | |
| SERIOUS ADVERSE Detail the symptoms if there is no diagnosis: EVENT: | | | | | | | SERIOUS CRITERIA □ PATIENT DIED (ENITUS) □ LIFE THREATENING | |
| DATE OF | KNOWLED | GE OF S | ERIOUS . | ADVERSE EV | VENT (DD/MM | I/YYYY): | ☐ HOSPITALIZATION ☐ PROLONGED HOSPIT | |
| | ION OF 1 | | | | ENT (Includi | ng relevant | ☐ PERSISTENCE OR SIG<br>DISABILITY/INCAPACH<br>☐ CLINICALLY RELEVA<br>☐ PREGNANCY | Y |
| | | | | | | | SEVERITY MILD MODERATE SEVERE LIFE THREATENING | |
| | | | | | | | ¿HAS THE SERIOU EVENT ENDED? | IS ADVERSE |
| PRODUCT | ? | QUALITY | Y BEEN | DETECTED | IN THE ST | JSPECTED | END DATE: | |
| ☐ YES ☐ NO IS IT A SUSPECTED TRANSMISSION OF AN INFECTIOUS AGENT THROUGH A MEDICAL PRODUCT?: ☐ YES ☐ NO | | | | | | | SAE OUTCOME: PERSISTENCE OF SAE RESOLVED WITHOUT SEQUELAE RESOLVED WITH SEQUELAE UNKNOWN EXITUS | |
| WAS THE SUBJECT WITHDRAWN FROM THE STUDY DUE TO THE SAE? ☐ YES ☐ NO | | | | | | | | |
| II. SUSPEC | I DRUG INFO | ORMATIC | ON | | | | | |
| SUSPECT | DRUG: | DAILY<br>(Include t | DOSE mits) | ROUTE | INDICATION<br>USE: | FOR | START DATE (dd/mm | ¥7777): |
| | AKEN WIT<br>Temporary is | | | - 7 | ion 🗆 Dose inci | rease 🗆 Dos | se decrease | |
| INTERRU | PTION DAT | E (dd/mm/) | ינינים): | | REINTR | ODUCTION | N DATE (dd/mm/yyyy): | |
| DID THE REACTION DIMINISH WHEN THE MEDICATION WAS SUSPENDED? WHEN THE ME WAS DECREAS | | | | | | TION DOSE WHEN THE MEDICATION WAS INTRUDUCED? | | The state of the s |
| ☐ YES | □ NO □ | NOTA | PPLY | | NO D NO | TADDIV | | □ NOT APPLY |

Page 1 de 2

Serious Adverse Evento Form Vs 3.0 de 01sep2020 - English Vs.



III. CONCOMITNANT MEDICATIONS AND MEDICAL HISTORY INDICATION CONCOMITANT DAILY ROUTE START END SAE MEDICATION DATE DOSE DATE (Include units) RELEVANT INFORMATION OF THE MEDICAL HISTORY (ej. Diagnostics, allergies, IV. RELATIONSHIP OF THE CAUSALITY OF THIS SERIOUS ADVERSE EVENT TO THE SUSPECTED DRUG/S
INVESTIGATOR'S JUDGMENT: SPONSOR'S JUDGMENT: ☐ Related ☐ Not related ☐ Not related ☐ Related V. INFORMATION OF THE SPONSOR AND INVESTIGATOR NAME AND PHONE OF THE INVESTIGATOR SPONSOR ADDRESS Fundación SEIMC-GESIDA WHO REPORT THE SAE: C/ Agustín de Betancourt nº 13 - entreplanta 28003 Madrid REPORT DATE (dd/mm/yyyy): COMPLEMENTARY REPORT ATTACHED ☐ YES ☐ NO INVESTIGATOR WHO COMPLETE THE REPORT: Name: Signature: \_\_\_ PERSONAL OF THE SPONSOR WHO RECEIVE THE REPORT: Name: Signature: \_ Reception date at SEIMC-GESIDA Foundation (DD/MM/YYYY): Page 2 de 2 Serious Adverse Evento Form Vs 3.0 de 01sep2020 - English Vs.

VOLVER Study protocol 4.0, 31 May 2021



#### **APPENDIX 5: PREGNANCY NOTIFICATION FORM**


| | Subject Identifier | Centre Number |
|---|---|---|
| REGNANCY NOTIFICATION | FORM | |
| This form should be completed accordin<br>Note: Most protocols do not require coll<br>Complete this form for each subject or subje<br>copy of the form to FSG (Email or fax numb | ection of subject's partner pregn<br>ect's partner who becomes pregnar | ancy. |
| Vho is this form being completed for, ✓ | one: Subject | |
| | Subject's partner | |
| NOTHER'S RELEVANT MEDICAL/FAMILY | Y HISTORY | |
| Nother's year of birth | Year | |
| Date of last menstrual period | Day Month Year | ] |
| estimated date of delivery | Day Month Year | ] |
| Was the mother using a method of contrace | eption? Yes No | |
| If Yes, specify: | | |
| Type of conception, ✓ one: | Normal (includes use | |
| Relevant laboratory tests and procedure | s (e.g., ultrasound, amniocentesis a | and chorionic villi sampling, |
| | s (e.g., ultrasound, amniocentesis a | and chorionic villi sampling, |
| | s (e.g., ultrasound, amniocentesis a | and chorionic villi sampling, |
| | s (e.g., ultrasound, amniocentesis a | and chorionic villi sampling, |
| ncluding dates of tests and procedures). | s (e.g., ultrasound, amniocentesis a | and chorionic villi sampling, |
| ncluding dates of tests and procedures). | Pre-term | |
| lumber of previous pregnancies | Pre-term | Full-term |
| lumber of previous pregnancies If applicable, record the number in the a | Pre-term ppropriate categories below: | Full-term |
| lumber of previous pregnancies If applicable, record the number in the a | ppropriate categories below: | Full-term |
| Number of previous pregnancies If applicable, record the number in the a | ppropriate categories below: Spontaneous abo Elective abortion Other | Full-term |
| Normal births Stillbirths Children born with defects | ppropriate categories below: Spontaneous abo Elective abortion Other | Full-term |

VOLVER Study protocol 4.0, 31 May 2021



| Protocol Identifier | | | | | Subject Ident | ifier | Centre Number | |
|---|---|---|---|---|---|---|---|---|
| DECHANOL | / NOTIFI | 0 A T/ | O | -0.044 | (O .: | | | |
| REGNANCY<br>ATHER'S RELE | | | | | 9 | ) | | |
| | | | | | | *** | | |
| Only recorded if re | | | | | | | | |
| Include habitual e<br>hromosomal disc | | | | | e abuse, chronic | c illnesses, far | nilial birth defe | ects/genetic/ |
| RUG EXPOSUR | ES | | | | | | | |
| n the following tab | nle list all m | edicatio | ne (inc | ludina eti | ıdv medications | ) the subject r | eceived durin | a the study |
| eriod (e.g. prescr | ription, OTC, | vaccin | es, reci | reational, | alcohol, etc.). E | nter the inve | stigational pi | roduct details |
| on the first line (i | | | | | | | | e). If there are |
| Drug Name | Route of | 3000 | | Started | Start Date | Stop Date | Ongoing | Reason for |
| (Trade Name | Admin. | Daily<br>Dose | | Pre-<br>Study | | otop Dato | Med-<br>ication | Medication |
| preferred) | For- | 2000 | | Judy | | | loution | |
| | maladon | | | Y=Yes | | | Y=Yes | |
| | | | | N=No | Day Month Year | Day Month Yea | | |
| | | <u> </u> | | | | | 37 | |
| | 50 | | | | | | 8 9 | |
| | 80 | | | | | | 30 31 | |
| Vas the subject w | ithdrawn from | n the s | tudy as | a result | of this pregnanc | y? 🗌 Ye | s No | |
| REPORTING INVI | ESTIGATOR | INFOR | RMATIC | ON (Forw | ard to a more a | opropriate phy | sician if need | ed) |
| lame | | | | | | | | |
| Address | | | | | | | | |
| City or State/Provi | | | | | | | | |
| Country | | | | | | | | |
| ost or Zip Code | | | | | | | | |
| elephone No | | | | | | | | |
| ax No | | | | | -8 | | | |
| nvestigator's sign | | | | | | Date | | onto Voss |
| confirming that th | e data on the | ese pag | es are | accurate | and complete) | | Day IVI | with redi- |
| nvestigator's nam | e (print) | | | | | | | |

Vs 1.0, date 25SEP2020.




# **APPENDIX 6: PREGNANCY FOLLOW-UP FORM**

| Protocol Identifier | Subject Identifier | Centre Number |
|---|---|---|
| REGNANCY FOLLOW-UP F | | |
| One form should be completed per foetus (e Who is this form being completed for, ✓ | E POST 16 | outu be completed for each twin |
| PREGNANCY STATUS | | |
| While pregnancy itself is not an AE or SAE<br>medical reasons will be recorded as an AE<br>considered to be an SAE and will be repor<br>result of a post-study pregnancy and cons<br>Investigator will be reported to FSG per th<br>information in former study participants, he | or SAE as described in the protocol. A<br>ted as described in the protocol. Furthe<br>idered reasonably related to the investi,<br>e protocol. Whilst the Investigator is not<br>s/she may learn of an SAE through spor | spontaneous abortion is alway:<br>ermore, any SAE occurring as a<br>gational product by the<br>t obligated to actively seek this |
| | | CATHODORNO TOTAL DE SECULOS |
| Stillbirth | Spontaneous | |
| Foetal death | Elective abo | rtion |
| Method used for delivery, specify_ | Other, specif | fy |
| <ul> <li>If male subject's partner is pregnan<br/>complete the information in the pap<br/>form.</li> </ul> | rm and on this paper Pregnancy Follow<br>t and the outcomes/associated events t<br>er SAE form and send together with th | fulfill the criteria of an SAE, ther<br>is paper Pregnancy Follow-up |
| section in the CRF. | 'associated events fulfil the criteria of a | n SAE, complete the SAE |
| FOETAL/NEONATAL STATUS | | |
| Normal | | |
| Birth defect (i.e., structural/chromo | somal disorder) Complete Serious Adv | erse Event pages |
| Other disorder (e.g., non-structura | , premature birth, intrauterine death/stil | llbirth) |
| If birth defects are diagnosed, is the origin | of the defect known? | No |
| If Yes, specify | | |
| INFANT INFORMATION | | |
| IN ANT IN CRIMATION | | |
| Date of birth/miscarriage/termination | Day Month | Year |
| Gestational weeks at birth/miscarriage/tern | nination Weeks | |
| Infant's sex | emale Unknown | |
| Length cm | Weight | g |
| Apgar score (0 - 10) First ass | essment Second | assessment |
| CONTRACTOR OF THE PROPERTY OF | CHARLEST TO THE RESIDENCE OF THE SECOND CONTROL OF THE SECOND CONT | Vs 1.0. date 25SEP20 |


| Prot | oco <mark>l Identifi</mark> | ier | | | Subject Ider | ntifier | Centre | Number |
|---|---|---|---|---|---|---|---|---|
| REGNANCY | TAILS (Provi | de addi | itional d | letails on | current labour/o | delivery/discharg | ge notes etc | ) |
| DRUG EXPOSUR<br>Complete drug sed<br>nclude drugs that | ction for all d | PREG | NANC<br>cluding | Y<br>i OTC/va | ccines) taken by | the mother dur | | |
| Drug Name<br>(Trade Name<br>preferred) | Route of<br>Admin.<br>or<br>For-<br>mulation | Total<br>Daily<br>Dose | Units | Started<br>Pre-<br>Study | Start Date | Stop Date | Ongoing<br>Med-<br>ication | Reason for<br>Medication |
| | | 2 - 3<br>K - 7 | | Y=Yes<br>N=No | Day Month Year | Day Month Year | Y=Yes<br>N=No | |
| | 38 | 8 8 | 8 | 2 | 3<br>5 | 20 7 | | |
| REPORTING INVI | ESTIGATOR | INFOR | RMATIC | N (Forwa | ard to a more ap | ppropriate physi | cian if neede | ed) |
| Name | | | | Title | _ Speciality _ | | | |
| Address | | | | | | | | |
| City or State/Provi | nce | | | | 8 | | | |
| Country | | | | | 2 | | | |
| ost or Zip Code_ | | | | | 2 | | | |
| elephone No | | | | | | | | |
| ax No | | | | | ş | | | |
| nvestigator's sign | ature<br>e data on the | ese pag | es are | accurate | and complete) | Date | Day M | onth Year |
| nvestigator's nam | e (print) | | | | | | | |

Vs 1.0, date 25SEP2020.



# **APPENDIX 7: LIVER EVENTS FORM**

Page


| Protocol Identifier | Site Identifier | Subject Identifier |
|---------------------|-----------------|--------------------|

# LIVER EVENT RECORD FOR INVESTIGATOR SPONSORED/VIIV SUPPORTED STUDIES

US:ENG (United States/English)

# COMPLETION GUIDELINES FOR CASE REPORT FORMS (CRFS)

#### GENERAL INSTRUCTIONS FOR CRF COMPLETION

- Complete CRFs in English; answer all questions on every page unless directed otherwise.
- Print neatly and legibly; use a black ballpoint pen and press firmly so that all copies are legible. Do not write information on page margins.
- Avoid use of abbreviations and acronyms whenever possible. If abbreviations must be used, use only clear abbreviations that are in standard medical use, or those supplied on instructional pages in this CRF. Enter Protocol and Subject Identifier in the space provided at the top of each CRF page.
- Do not write the Subject's name or initials anywhere inside the CRF. Record all values in the units indicated on the CRF.
- Where boxes are provided in the CRF to record numbers, complete as follows, using leading zeroes if necessary: 6 recorded as  $\boxed{0}$   $\boxed{6}$ .
- Ensure that information classified as "Other, specify" does not fit into one of the listed categories. Record a oncise reason in the "specify" field that accompanies "Other" if "Other" is \( \structure{\chi} \).

  If extra pages need to be inserted between numbered CRF pages, do the following: insert the first extra page
- after the last numbered page in the section of the CRF affected (e.g., Concomitant Medications) and number the extra page as nn.01. Subsequent extra pages are then numbered nn.02, nn.03 etc.

# MISSING INFORMATION

- Use the following abbreviations for missing information.
  - not available/not applicable
  - ND not done unknown
  - · NR no result (to be used only for missing data recorded on Local Lab pages)

#### CRF CORRECTION PROCESS

- . Draw a single line through an incorrect entry and write the correct information nearby.
- Initial and date all corrections, additions or deletions.
- DO NOT erase, write over, use correction fluid or tape, or re-copy the original page to correct errors.



|---------------------|
| Protocol Identifier |

# **ACTION IS REQUIRED**

# LIVER EVENT RECORD (INVESTIGATOR SPONSORED/VIIV SUPPORTED STUDIES) INVESTIGATOR INSTRUCTIONS

Liver Event Record Completion
 Complete this Liver Event Record for all possible, suspected, implied, and/or probable cases of liver event.
 For serious adverse events (SAE), please ensure data provided here is consistent with the SAE CRF. If the

Inform Fundación SEIMC-GESIDA

Mail or fay (fay preferred) the completed Liver Event Record

SAE CRF is updated, please resubmit to FSG.

Mail or fax (fax preferred) the completed Liver Event Record within one week of the clinical assessment for liver event to GlaxoSmithKline.

Retain a copy of the Liver Event Record for your files.

Attention: Fundación SEIMC-GESIDA C/Agustín de Betancourt, 13 Entreplanta 28003 Madrid

FAX: +34 91 554 22 83



US:ENG (United States/English)


| Protoc | ol Identifier Subje | ct Identifier |
|---|---|---|
| NVESTIGATOR INFORMAT | SORED/VIIV SUPPORTED STUDIES, | i |
| Print clearly. | | |
| Investigator's Name | | |
| Site Number | | |
| Investigator's Address | | (Institution) |
| | | (Internal Address) |
| | | (Street Address) |
| | | (City, State, Province<br>Postal Code) |
| | | (Country) |
| Investigator's Telephone Number | | |




| Protocol Identifier | Site Identifier | Subject Identifier | Visit Date Day Month Year |
|---|---|---|---|

# LIVER EVENTS

| | sample collection which resulted in the subject meeting protocol<br>e a scheduled sample collection, so this "Visit Date" may be the same |
|---|---|
| Which liver chemistry result reached or exce criteria? ✓ all that apply | eded protocol-defined investigational product stopping/interruption |
| [1] ALT (alanine aminotransferase) | |
| [3] Total bilirubin | |
| [7] Direct bilirubin | |
| [8] INR | |
| [OT] Other | |
| When did the liver event occur? | |
| [D] During the treatment period | |
| [A] After the treatment period | |
| If the liver event occurred during treatment p<br>treatment period. | period record start and stop date of investigational product for that |
| If the liver event occurred after treatment pe<br>recent period prior to the liver event. | riod record start and stop date of investigational product for the most |
| Start date of Investigational Product Da | y Month Year |
| End date of Investigational Product Day | y Month Year |

Vs 1.0, date 25SEP2020.




| Protocol Identifier | Subject Identifier |
|---|---|
| Protocol identifier | |
| .IVER EVENTS (Continued) | |
| Record the details of any Adverse Events or exacerbations of A<br>Form OR the Serious Adverse Event Form. Exacerbations of A<br>severity. | |
| It is particularly important to record any significant hypotension<br>elevation.<br>It is particularly important to record any gallbladder or biliary di<br>study. | 7.F |
| Is the subject age 55 or older? | |
| [Y] Yes [M] No | |
| If female, is the subject pregnant? | |
| [Y] Yos [N] No [X] Not applicable | |
| If Yes, ensure Pregnancy Notification Form has been comp | leted. |
| Were any diagnostic imaging tests of the liver or hepatobiliary<br>computerized tomography or CAT scan, magnetic resonance in<br>cholangiopancreatography, or other)? | |
| [Y] Yos [N] No | |
| If Yes, were the results normal? | |
| [Y] Yes [N] No | |
| If No, record the details on the Imaging form. Ensure the ov<br>the Non-Serious Adverse Event form or Serious Adverse E | |
| Were any liver biopsies performed? | |
| [Y] Yos [N] No | |
| If Yes, complete Liver Biopsy form. | |
| Does the subject use herbals, complementary or alternative modrugs? | edicines, food supplements (vitamins) or illicit |
| [Y] Yes [N] No | |

Vs 1.0, date 25SEP2020.

If Yes, record on the appropriate Concomitant Medication form. Did the subject fast or undergo significant dietary change in the past week?

[Y] Yos [N] No



|---------------------|
| Protocol Identifier |

# LIVER EVENTS

# DEFINITIONS

# CURRENT MEDICAL CONDITIONS

Conditions from which the subject is currently suffering, regardless of how long they have been present. If the subject has had a recurring condition that is not present at the time of the assessment, it can be classed as current if, in the Investigator's opinion it is likely to recur during the study.

#### PAST MEDICAL CONDITIONS

Conditions from which the subject has suffered in the past, but are no longer present. A past condition may have stopped as recently as the day prior to being assessed.

NO MEDICAL CONDITION

No current or past condition.

Vs 1.0, date 25SEP2020.

#### ALCOHOL INTAKE AT ONSET OF LIVER EVENT INVESTIGATOR INSTRUCTIONS

ALCOHOL CONVERTER

1 unit of alcohol in US = 1.5oz hard liquor, 1 beer, 4oz wine

1 unit of alcohol in UK = 1 measure of spirits, 1/2 pint beer, 1 small glass of wine (125ml)

Vs 1.0, date 25SEP2020.




| | Subject Identifier | | |
|---|---|---|---|
| - 8 | , A. | | |
| Current | Past | No Medical Con | dition |
| [1] | [2] | [5] | |
| | 8 2 | | |
| 15 | 8 8 | | |
| 92 | 0 3 | | |
| 102 | 0 0 | | |
| | 8 8 | | |
| 10 | | | |
| 100 | | | |
| | 60 20<br>60 00 | | |
| | 0 9 | | |
| | R 91 | | |
| 3 | 65 /9 | | |
| including In | vestigatio | nal Product) | |
| * | 68 88 | | |
| 12 | Current | Past | |
| esponse for | 191 | [2] | |
| | 0 0 | | |
| | 10 93 | | |
| Current<br>[1] | Past<br>[2] | No Medical Con<br>[5] | dition |
| 90 | 0 3 | | |
| | 8 8 | | |
| 100 | | | |
| | 9 9 | | |
| | K 3 | | |
| 18 | k 3 | | |
| | s including In | s including Investigation Current [1] | s including Investigational Product) response for |




| 00 | SAL | _ | - | _ | MT | 1 4 1 |
|----|-----|---|---|---|----|-------|

| Protocol Identifier | Site Identifier | Subject Identifier |
|---|---|---|
| IVER EVENT RECORD<br>INVESTIGATOR SPONSOREI | D/VIIV SUPPORTED S | TUDIES) (Continued) |
| Provide a textual description of the liver ever<br>interruptions of liver therapy including dates<br>contributing factors, alternative etiologies, a<br>For serious AE (SAE), please use the SAE<br>resubmit to GSK. | t, treatment required to stabilize the<br>and any other relevant information | he reaction, resolution/outcome, other<br>n. Use additional pages as needed. |
| S:ENG (United States/English) IVER EVENT RECORD INVESTIGATOR SPONSORE INVESTIGATOR'S SIGNATURE | D/ViiV SUPPORTED S | TUDIES) (Continued) |
| The Investigator is accountable for this data to a medically qualified Sub-investigator. | a. However, the Principal Investig | ator may delegate signature authority |
| confirm that I have reviewed the data in the colleagues is, to the best of my knowledge, | | |
| Investigator's Signature: | | Date Day Month Year |
| Investigator's Name (print)<br>S:ENG (United States/English) | | |



# **APPENDIX 8: LIVER EVENTS BIOPSY FORM**

|---------------------|-----------------|--------------------|
| Protocol Identifier | Site Identifier | Subject Identifier |

# LIVER EVENT BIOPSY RECORD FOR INVESTIGATOR SPONSORED/VIIV SUPPORTED STUDIES

US:ENG (United States/English)

# COMPLETION GUIDELINES FOR CASE REPORT FORMS (CRFS)

#### GENERAL INSTRUCTIONS FOR CRF COMPLETION

- Complete CRFs in English; answer all questions on every page unless directed otherwise.
   Print neatly and legibly; use a black ballpoint pen and press firmly so that all copies are legible.
- Do not write information on page margins.
- Avoid use of abbreviations and acronyms whenever possible. If abbreviations must be used, use only clear abbreviations that are in standard medical use, or those supplied on instructional pages in this CRF.
- Enter Protocol and Subject Identifier in the space provided at the top of each CRF page.
- Do not write the Subject's name or initials anywhere inside the CRF.
   Record all values in the units indicated on the CRF.
- · Where boxes are provided in the CRF to record numbers, complete as follows, using leading zeroes if necessary: 6 recorded as 0 6.
- Ensure that information classified as "Other, specify" does not fit into one of the listed categories. Record a
  concise reason in the "specify" field that accompanies "Other", if "Other" is 

  √.
- If extra pages need to be inserted between numbered CRF pages, do the following: insert the first extra page after the last numbered page in the section of the CRF affected (e.g., Concomitant Medications) and number the extra page as nn.01. Subsequent extra pages are then numbered nn.02, nn.03 etc.

#### MISSING INFORMATION

- Use the following abbreviations for missing information.
- NA not available/not applicable · ND
- not done
- UNK unknown
   NR no result
- no result (to be used only for missing data recorded on Local Lab pages)

#### CRF CORRECTION PROCESS

- Draw a single line through an incorrect entry and write the correct information nearby.
- Initial and date all corrections, additions or deletions.
- DO NOT erase, write over, use correction fluid or tape, or re-copy the original page to correct errors.




|---------------------|
| Protocol Identifier |

# **ACTION IS REQUIRED**

# LIVER EVENT BIOPSY RECORD (INVESTIGATOR SPONSORED/VIIV SUPPORTED STUDIES) INVESTIGATOR INSTRUCTIONS

# 1. Liver Event Biopsy Record Completion

Complete this Liver Event Biopsy Record for all possible, suspected, implied, and/or probable cases of liver event biopsy.

For serious adverse events (SAE), please ensure data provided here is consistent with the SAE CRF. If the SAE CRF is updated, please resubmit to FSG.

#### 2. Inform GlaxoSmithKline

Mail or fax (fax preferred) the completed Liver Event Biopsy Record within one week of the clinical assessment for liver event biopsy to GlaxoSmithKline.

Retain a copy of the Liver Event Biopsy Record for your files.

Attention:Fundación SEIMC-GESIDA

C/ Agustín de Betancourt, 13-Entreplanta 28003 - Madrid

FAX: +34 91 554 22 83



| Protocol Identifier | Site Identifier | Subject Identifier |
|---|---|---|
| Protocoridentiner | | <del>, , </del> |
| IVER EVENT BIOPSY F | RECORD | |
| INVESTIGATOR SPONS | SORED/VIIV SUPPORTED STUDIES | ) |
| Print clearly. | ion | |
| 5.48.30=77=370 <b>=</b> 250 | | |
| Investigator's Name | | |
| Site Number | | |
| Investigator's Address | | (Institution) |
| | | (Internal Address) |
| | | (Street Address) |
| | | (City, State, Province<br>Postal Code) |
| | | (Country) |
| Investigator's Telephone Number | | |




| Protocol Identifier | Site Identifier | Subject Identifier |
|---------------------|-----------------|--------------------|

| Complete a separate form for each liver biopsy perfor | rmed. |
|---|---|
| Date of liver biopsy | |
| Day Month | year |
| Approximate size of liver biopsy mm (num | ber from 0 - 50) |
| A. Final Diagnosis ✓ all that apply: | |
| [A0] Normal | [A 1 6] Alcoholic hepatitis |
| [A1] Acute hepatitis | [A 1 7] Hepatic granulomas |
| [A2] Chronic hepatitis | [A 1 8] Sarcoidosis |
| [A3] Cholestatic hepatitis | [A 1 9] Fibrosis |
| [A4] Drug-induced cholestasis | [A 20] Cirrhosis |
| [A5] Acute viral hepatitis | [A 21] Primary biliary cirrhosis |
| [A6] Chronic viral hepatitis | [A 2 2] Primary sclerosing cholangitis |
| [A7] Drug-induced hepatitis | [A 2 3] Autoimmune overlap syndrome |
| [A8] Autoimmune hepatitis | [A 2 4] Hemochromatosis |
| [A9] Bridging necrosis | [A 2 5] Alpha-1-antitrypsin deficiency |
| A 1 0] Submassive hepatic necrosis | [A 2 6] Wilson's disease |
| A 11] Massive hepatic necrosis | [A 27] Veno-occlusive disease |
| A 1 2] Steatosis - microvesicular | [A 2 8] Budd-Chiari syndrome |
| A 1 3] Steatosis - macrovesicular | [A 2 9] Neoplasia |
| A 1 4] Steatosis - mixed | [A 9 9] Other, specify: |
| A 15] Non-alcoholic steatohepatitis | |
| 3. Liver Architecture ✓ all that apply: | |
| [B1] Normal | [B13] Interface hepatitis (periportal hepatitis or |
| [R 2] Bridging fibrosis | piecemeal necrosis) |
| [B3] Diffuse fibrosis | [B14] Ischaemic necrosis |
| [84] Nodular regenerative hyperplasia | [B15] Centrolobular (Zone 3) necrosis |
| [85] Congenital hepatic fibrosis | [816] Focal coagulative necrosis |
| [86] Cirrhosis | [B17] Centrolobular (Zone 3) coagulative |
| [87] Centrilobular congestion | necrosis |
| [R8] Endophlebitis | [B18] Bridging hepatocellular necrosis |
| [R 9] Veno-occlusive disease | [819] Massive or panlobular hepatocellular |
| B 1 0] Canalicular cholestasis | necrosis |
| B11] Apoptosis | [B20] Dysplasia |
| B 1 2] Focal (or spotty or mild) hepatocellular | [B 21] Neoplasia |
| necrosis | [B99] Other, specify: |




| Protocol Identifier | Site Identifier | Subject Identifier |
|---------------------|-----------------|--------------------|

| C. Description of Liv | er Cells or Hepatocytes ✓ all that | apply: | |
|---|---|---|---|
| [Co] Normal | | [C3] | Pseudoxanthomatous |
| [C1] Ballooning | | [C4] | Multinucleated giant hepatocytes |
| [C2] Acidophilic | | [C 9 9] | Other, specify: |
| D. Liver Cell or Hepa | tocyte Inclusions or Vacuoles ✓ | all that appl | y: |
| [D0] No inclusion | ns | [88] | "Ground Glass" inclusions |
| [D1] Macrovesic | ular steatosis | [60] | Lipofuscin pigment |
| [D 2] Microvesicu | ular steatosis | [D10] | Hemosiderin granules |
| [D3] Bile accum | ulation | [D11] | Orcein-positive cytoplasmin granules |
| [D4] Diastase-re | sistant, PAS-positive cytoplasmic | [D12] | Protoporphyrin crystals (birefringent under<br>polarised light) |
| | titrypsin inclusions | [013] | Uroporphyrin crystals (red fluorescence |
| [D6] Megamitoc | | 197.91 | under ultraviolet light) |
| [D7] Mallory boo | | [099] | Other, specify: |
| . Hepatocyte or Live | er Cell Nuclear Abnormalities 🗸 | all that apply | |
| [Fo] None | | [E 4] | HSV inclusions |
| [E1] Hepatocellu | ular <mark>m</mark> itoses | [E 5] | Varicella inclusions |
| | d or multinucleated hepatocytes | [E 9 9] | Other, specify: |
| [F3] CMV inclus | ion bodies | | |
| Liver or Lobular In | filtrates ✓ all that apply: | | |
| [F0] None | | [F 5] | Macrophages and proliferating Kupffer |
| [F1] Eosinophils | | | cells |
| [F2] Lymphocyte | es | [F6] | Granulomas |
| [F3] Plasma cell | ls | [F99] | Other, specify: |
| [F4] Neutrophils | | | |
| 3. Portal Tract Inflam | nmation ✓ all that apply: | | |
| [G0] None | | [G4] | Neutrophils |
| [G1] Eosinophils | k | [G5] | Histocytes and macrophages |
| [G2] Lymphoid a | ggregates and/or follicles | [G99] | Other, specify: |
| [G3] Plasma cell | s | | |




| Protocol Identifier | Site Identifier | Subject Identifier |
|---|---|---|
| IVER BIOPSY (Continued) | | |
| I. Bile Ducts ✓ all that apply: | | |
| [Ho] Normal | [H3] Pauci | ty of bile ducts |
| [H1] Proliferation of bile ducts (bile ductula | [H4] Peridu | uctal fibrosis |
| reaction) | | , specify: |
| [H2] Dilation, degeneration or disruption of bile ducts | portal | |
| . Portal Veins ✓all that apply: | | |
| [10] Normal | [13] Neopl | astic invasion of portal vein |
| [11] Pyelophlebitis | | lomatous compression of portal vei |
| [12] Thrombosis, sclerosis or occlusion of | portal [199] Other, | specify: |
| vein | | |
| J. Liver Infections ✓ all that apply: | | |
| [Jo] Normal | [J5] Histop | olasma capsulatum |
| [J1] Leishmaniasis donovani | | pacterium tuberculosis |
| [J2] Plasmodium falciparum | [J7] Other | mycobacterial species |
| [J3] Toxoplasmosis | [J99] Other | , specify: |
| [J4] Cryptococcus neoformans | | |
| <ol> <li>Parasites or Ova ✓ all that apply:</li> </ol> | | |
| [K0] None | [K 4] Echine | ococcus cysts |
| [K1] Schistosome and/or ova | [K 5] Hepat | ic capillariasis worms and/or ova |
| [K2] Ascaris and/or ova | [K 9 9] Other | specify: |
| [K3] Toxocara and/or ova | | |
| Histologic Staining or Additional Studies O | Obtained 🗸 all that apply: | |
| [L1] Haematoxylin and eosin (or H & E) | [L10] Rhoda | anine (copper) |
| [L2] Masson | | anic acid (copper) |
| [L3] Toluidine blue or Giemsa | [L 1 2] Orcein | n, aldehyde fuchsin or Victoria blue |
| [L4] Prussian blue | | on microscopy |
| [L5] Periodic Acidic Schiff (PAS), with or w | ithout [L14] Hepat | itis A immunostains positive |
| diastase | [L15] Hepat | itis B core antigen or hepatitis B |
| [L6] Oil red O | surfac | ce antibody immunostains positive |

[L 1 6] Hepatitis D immunostains
[L 1 7] Other immunostains
[L 9 9] Other, specify:

Vs 1.0, date 25SEP2020.

[L7] Congo red
[L8] Hall's stain
[L9] Gridley's stain




| Protocol Identifier | Site Identifier | Subject Identifier |
|---|---|---|
| VER EVENT BIOPSY REC<br>NVESTIGATOR SPONSORI<br>ARRATIVE/COMMENTS | | TUDIES) (Continued) |
| rovide a textual description of the liver e<br>ny/all interruptions of liver therapy inclu-<br>utcome, other contributing factors, alter<br>ages as needed. | ding dates, treatment required to st | abilize the reaction, resolution/ |
| or serious AE (SAE), please use the SA<br>submit to FSG. | E CRF for narrative description. If | the SAE CRF is updated, please |
| :ENG (United States/English) | | |

# LIVER EVENT BIOPSY RECORD (INVESTIGATOR SPONSORED/ViiV SUPPORTED STUDIES) (Continued) INVESTIGATOR'S SIGNATURE

| The Investigator is accountable for this data. However, the Princip | al Investigator m | ay delega | ate signat | ure authori |
|---|---|---|---|---|
| to a medically qualified Sub-investigator. | | | | |
| I confirm that I have reviewed the data in this report for this subject | t. All information | entered | by myself | or my |
| colleagues is, to the best of my knowledge, complete and accurat | e, as of the date | below. | storetiset. | 2010-00-00 |
| colleagues is, to the best of my knowledge, complete and accurate investigator's Signature: | e, as of the date | Day | Month | Year |

Ve 1.0; date 258EP2020.



# APPENDIX 9: POSSIBLE SUICIDALITY-RELATED ADVERSE EVENT FORM

| cor | NFIDENTIAL | |
|---------------------|-----------------|--------------------|
| Protocol Identifier | Site Identifier | Subject Identifier |

# POSSIBLE SUICIDALITY-RELATED ADVERSE EVENT FOR INVESTIGATOR SPONSORED/VIIV SUPPORTED STUDIES

US:ENG (United States/English)

# POSSIBLE SUICIDALITY-RELATED ADVERSE EVENT

INSTRUCTIONS FOR COMPLETING POSSIBLE SUICIDALITY-RELATED ADVERSE EVENT FORMS

Complete the "Possible Suicidality-Related Adverse Event" CRF Form if there is an occurrence of an adverse event which, in the investigator's judgement, is a possible suicidality-related event. This may include, but is not limited to, an event that involves suicidal ideation, a preparatory act toward imminent suicidal behaviour, a suicide attempt, or a completed suicide.

The event must also be reported on the Serious Adverse Events (SAE) CRF using the same terminology. Please ensure data provided here is consistent with the SAE CRF.



# CONFIDENTIAL Protocol Identifier

#### COMPLETION GUIDELINES FOR CASE REPORT FORMS (CRFS)

#### GENERAL INSTRUCTIONS FOR CRF COMPLETION

- Complete CRFs in English; answer all questions on every page unless directed otherwise.
- Print neatly and legibly; use a black ballpoint pen and press firmly so that all copies are legible.
- · Do not write information on page margins.
- Avoid use of abbreviations and acronyms whenever possible. If abbreviations must be used, use only clear abbreviations that are in standard medical use, or those supplied on instructional pages in this CRF.

  Enter Protocol and Subject Identifier in the space provided at the top of each CRF page.
- Do not write the Subject's name or initials anywhere inside the CRF.
- Record all values in the units indicated on the CRF.
- Where boxes are provided in the CRF to record numbers, complete as follows, using leading zeroes if necessary: 6 recorded as 0 | 6 |.
- Ensure that information classified as "Other, specify" does not fit into one of the listed categories. Record a
- concise reason in the "specify" field that accompanies "Other", if "Other" is  $\checkmark$ . If extra pages need to be inserted between numbered CRF pages, do the following: insert the first extra page after the last numbered page in the section of the CRF affected (e.g., Concomitant Medications) and number the extra page as nn.01. Subsequent extra pages are then numbered nn.02, nn.03 etc.

#### MISSING INFORMATION

- Use the following abbreviations for missing information.
  - · NA · ND not available/not applicable
  - not done
  - UNK unknown
- no result (to be used only for missing data recorded on Local Lab pages)

#### CRF CORRECTION PROCESS

- Draw a single line through an incorrect entry and write the correct information nearby.
- Initial and date all corrections, additions or deletions.
- DO NOT erase, write over, use correction fluid or tape, or re-copy the original page to correct errors.



| | C | ONF | IDEN | TIAL |
|---------------------|---|-----|------|------|
| Protocol Identifier | | | | |

#### **ACTION IS REQUIRED**

# POSSIBLE SUICIDALITY-RELATED ADVERSE EVENT RECORD (INVESTIGATOR SPONSORED/VIIV SUPPORTED STUDIES) INVESTIGATOR INSTRUCTIONS

Mail or fax (fax preferred) the completed Possible Suicidality-Related Adverse Event Record within one week of the clinical assessment for Possible Suicidality-Related Adverse Event to Fundación SEIMC-GESIDA.

Retain a copy of the Possible Suicidality-Related Adverse Event Record for your files.

Attention: Fundación SEIMC-GESIDA C/ Agustín de Betancourt nº 13 - entreplanta Madrid 28003

Fax: +34 915542283

US:ENG (United States/English)


| Protocol Identifier | Site Identifier | Subject Identifier |
|---------------------|-----------------|--------------------|

# POSSIBLE SUICIDALITY-RELATED ADVERSE EVENT RECORD (INVESTIGATOR SPONSORED/VIIV SUPPORTED STUDIES) INVESTIGATOR INFORMATION

| Print clearly. | |
|---------------------------------|-----------------------------------------|
| Investigator's Name | |
| Site Number | |
| Investigator's Address | (Institution) |
| | <br>(Internal Address) |
| | <br>(Street Address) |
| | (City, State, Province,<br>Postal Code) |
| | (Country) |
| Investigator's Telephone Number | |
| Investigator's E-Mail Address | |




| Protocol Identifier | | 5 | Subject Identifier |
|---|---|---|---|
| POSSIBLE SUICIDALITY-RE | LATED ADVERSE EVEN | IT | |
| SECTION 1 | secons was | | 2000 100 200 |
| | | sessed by the investigator during the study | |
| Note: Review SAE CRF pages aiready | | on is available, update and resubmit the | |
| | Event | | Start Date Day Month Year |
| | e.g., Fleeting suicidal thoughts | | 25 Jan 14 |
| | 500 St 550 | | 5 S |
| | | | 5 k |
| | | | 0 |
| | | | 2.5 |
| SECTION 2 Possible Cause(s) of Pos | sible Suicidality-related Adverse E | Event: | -15 |
| Disease under study [Y] | Yos [N] No | Withdrawal of study treatment(s) | [Y] Yes [N] No |
| Concomitant medication(s) [Y]<br>Record in Section 8 | Yos [N] No | Study treatment dose change | [Y] Yos [N] No |
| Comorbid psychiatric condition(s) [Y]<br>Record in Section 8 | Yos [N] No | Lack of efficacy | [Y] Yos [N] No |
| Medical condition(s) [Y]<br>Record in Section 8 | Yes [N] No | Study treatment(s) | [Y] Yes [N] No |
| Psycho-social stressors [Y] Record in Section 5 15:FMG (United States/Fnolish) | Yos [N] No | Other, specify | |
| | Protocol Identifier | NFIDENTIAL | |
| | | | Subject Identifier |
| POSSIBLE SUICIDALITY-RE | I ATED ADVERSE EVE | NT (Continued) | |
| SECTION 3 Provide this information, | | | |
| | | If Yes, provide information: | |
| <ol> <li>Has the subject had any psychiatric<br/>conditions in the past?</li> </ol> | [Y] Yes [N] No | ii res, provide iiromason. | |
| Has the subject had any suicidal | [Y] Yes [N] No | If Yes, provide information: | |
| ideation, behaviour or self-harm in | | | |
| the past? | | | |
| 3. Subject's current use of illicit drugs? | [Y] Yes [N] No | If Yes, provide information, in has been obtained: | ncluding results of a drug screen test if one |
| | 3. | | |
| Subject's current use of alcohol? | [Y] Yes [N] No | If Yes, provide information, in<br>has been obtained: | cluding results of an alcohol level test if on |
| 5. Family history of suicidality? | [Y] Yes [N] No [U] | Unk If Yes, provide information: | |
| | 1 200 mm 1 100 mm 1 100 mm | 1 1 1 1 1 1 1 1 1 1 1 1 1 1 1 1 1 1 1 1 | |
| <ol><li>Family history of psychiatric<br/>disorders?</li></ol> | [Y] Yes [N] No [U] | Unk | |
| 0.50.40.31 | | | |
| | J. | | |




| Protocol Identifier | Subject Identifier |
|---|---|
| OSSIBLE SUICIDALITY-RELATED ADVERSE EVENT (Co | |
| SECTION 4 Provide information on the subject's current psycho-social stressor<br>inances, stress, etc. | rs. For example, isolation, problems with family, relationships, work, |
| SECTION 5 Provide information on any relevant and/or recent suicidal ideation,<br>nvestigator, for this index event i.e., provide details, including any suicidal thoughts | |
| he subject acting upon these thoughts. | |
| :ENG (United States/English) | |
| 2212221 | |
| CONFIDENT | IAL |
| Protocol Identifier | Subject Identifier |
| OSSIBLE SUICIDALITY-RELATED ADVERSE EVENT (Co | |
| SECTION 6 Provide information on any suicidal behaviour present during the | study, as assessed by the investigator, for this index event, i.e. |
| Details of any suicidal behaviour, including any plan, preparations, and/or attempt | |
| Description of the associated frequency, severity and duration of these behaviour | 5 |
| Likelihood of the subject acting upon plans and preparations | |
| If possible, description of the subject's intent (or evidence of attention seeking be | haviour\ |
| | naviour) |
| Description of the degree of impulsivity or premeditation | |
| Description of the subject's mood and thoughts before and after the behaviour | |
| SECTION 7 Provide any additional comments or explanation, including, | nited to, both medical and psychiatric treatment, outcome and |
| ollow-up. | 100 |
| S:ENG (United States/English) | |



|---------------------|
| Protocol Identifier |

# POSSIBLE SUICIDALITY-RELATED ADVERSE EVENT RECORD (INVESTIGATOR SPONSORED/VIIV SUPPORTED STUDIES) (Continued) INVESTIGATOR'S SIGNATURE INVESTIGATOR INSTRUCTIONS

The Investigator is accountable for this data. However, the Principal Investigator may delegate signature authority to a medically qualified Sub-investigator.

| I confirm that I have reviewed the data in this report for this subject. All in<br>colleagues is, to the best of my knowledge, complete and accurate, as of | | | d by myself | or my |
|---|---|---|---|---|
| Investigator's Signature: | Date | Day | Month | Year |
| Investigator's Name (print) | | -55% | | |



# **APPENDIX 10: LIVER IMAGING RECORD**

| | | Page |
|---------------------|-----------------|--------------------|
| Protocol identifier | Site Identifier | Subject Identifier |

# LIVER IMAGING RECORD FOR INVESTIGATOR SPONSORED/ViiV SUPPORTED STUDIES

US:ENG (Linted States/English)

# COMPLETION GUIDELINES FOR CASE REPORT FORMS (CRFS)

#### GENERAL INSTRUCTIONS FOR CRF COMPLETION

- Complete CRFs in English; answer all questions on every page unless directed otherwise.
   Print neatly and legibly; use a black balipoint pen and press firmly so that all copies are legible.
- Do not write information on page margins.
- Avoid use of abbreviations and acronyms whenever possible. If abbreviations must be used, use only clear
- abbreviations that are in standard medical use, or those supplied on instructional pages in this CRF. Enter Protocol and Subject identifier in the space provided at the top of each CRF page.
- Do not write the Subject's name or initials anywhere inside the CRF.
- Record all values in the units indicated on the CRF.
- Where boxes are provided in the CRF to record numbers, complete as follows, using leading zeroes if necessary: 6 recorded as 0 0
- If extra pages need to be inserted between numbered CRF pages, do the following: insert the first extra page after the last numbered page in the section of the CRF affected (e.g., Concomitant Medications) and number the extra page as nn.01. Subsequent extra pages are then numbered nn.02, nn.03 etc.

## MISSING INFORMATION

- Use the following abbreviations for missing information.
  - not available/not applicable
  - · ND not done
  - UNK unknown
     no result
    - no result (to be used only for missing data recorded on Local Lab pages)

#### CRF CORRECTION PROCESS

- Draw a single line through an incorrect entry and write the correct information nearby.
- initial and date all corrections, additions or deletions.
- DO NOT erase, write over, use correction fluid or tape, or re-copy the original page to correct errors.



| | 16 | CONF | IDEN | CHAL |
|---------------------|----|------|------|------|
| Protocol Identifier | | | I | |

# **ACTION IS REQUIRED**

# LIVER IMAGING RECORD (INVESTIGATOR SPONSORED/ViiV SUPPORTED STUDIES) INVESTIGATOR INSTRUCTIONS

1. Liver imaging Record Completion

Complete this Liver imaging Record for all possible, suspected, implied, and/or probable cases of liver imaging.

For serious adverse events (SAE), please ensure data provided here is consistent with the SAE CRF. If the SAE CRF is updated, please resubmit to FSG.

2. Inform Fundación SEIMC-GESIDA

Mail or fax (fax preferred) the completed Liver imaging Record within one week of the clinical assessment for liver imaging to Fundación SEIMC-GESIDA.

Retain a copy of the Liver imaging Record for your files.

Attention: Fundación SEIMC-GESIDA

C/Agustín de Betancourt, 13 - Entreplanta 28003 Madrid

FAX: +34 91 554 22 83




| Protocol identifier | Subject identifier |
|---------------------|--------------------|

# LIVER IMAGING RECORD (INVESTIGATOR SPONSORED/ViiV SUPPORTED STUDIES)

| Print clearly. | |
|--------------------------------|-----------------------------------------|
| invesägator's Name | |
| Site Number | |
| nvestigator's Address | (Institution) |
| | (Internal Address) |
| | (Street Address) |
| | (City, State, Province,<br>Postal Code) |
| | (Country) |
| nvestigator's Telephone Number | |
| nvestigator's E-Mail Address | |



| Protocol identifier | Site identifier | Subject identifier |
|---|---|---|
| IVER IMAGING | | 22 |
| Complete a separate form for each individual in | naging test performed. | |
| Date of hepatic or liver imaging test Day | March Veet | |
| What method was used for this imaging test<br>a separate form for each test). | ? ✓one: (If more than one in | naging test was performed, complet |
| 1) Utrasound - transabdominal | (e) Postron ( | Emission Tomography (PET) |
| 변 Ultrasound - endoscopic | | Emission Tomography/Computed |
| (8) Magnetic Resonance Imaging (MRI) | Tomogray | ony (PET/CT) |
| 4] Computerised Tomography (CT) | [UT] Other, sp | ecify: |
| 5] Endoscopic Retrograde | | |
| Cholangiopancreatography (ERCP) | | |
| Are images technically adequate? ✓ one: | | |
| VI Optimal | [8] Not read: | sole |
| 리 Readable, but not optimal | [OT] Other, sp | ecify: |
| A. Indicate the liver size Jone: | | |
| A1 Normal size | (A 4) Segmen | ital hypertrophy |
| A 2 I Hypertrophy (or enlarged) | | pecify: |
| A 31 Atrophy (or smaller than normal) | | |
| B. Indicate the liver texture ✓one | | |
| | - · · · | TO RESONATE MESSAGES |
| B1 Normal | | or suggestive of cirrhosis pecify: |
| B2 Heterogeneous<br> B3 Suggestive of fibrosis | (AAMILLI OMB, S | pecity. |
| | value v rought | |
| C. Grade the diffuse and/or geographic fatty | inflitrate of the liver / one | |
| C1] Not applicable - no fatty infitration | IC4 Severe | |
| C21 Mild (≤25%) | (C98) Other, s | pecify: |
| C 3] Moderate (>25% to <75%) | | |
| D. Asoltes present √one: | | |
| D1) None present | [Dist] Yes - m | oderate or severe amount |
| D2I Ves - small amount | 1 ( S 2 ( S 2 ) 1 ( S 2 ) | pecify: |




| | Protocol Identifier 81 | bjeat identifier |
|---|---|---|
| _ | | |
| | IMAGING (Continued) | 0.0000000000000000000000000000000000000 |
| E. Are F | coal Hepatic Lesions characterisable? | fall that apply: |
| E 85 | Not applicable - no hepatic lesions | E S Hemangloma |
| E 1] | Solid | Focal Nodular Hyperplasia |
| [2] | Cystic | [E99] Other, specify: |
| Galle | tones or galibladder lesions? ✓ all that a | ng/v: |
| F 08 | | |
| | None | |
| F11_ | Galistones | [Fit] Cholecystits |
| F 25 | Galibladder polyp(s) | F 7 ☐ Galibladder wall calcfication |
| | Sludge | F 0 Gallbladder mass |
| F4] | Galibladder wall thickening/oedema | [F99] Other, specify: |
| 3. Billar | y duotal lecions? ✓all that apply: | |
| 0.05 | None | [04] Acute Cholangitis |
| 01] | Intrahepatic ductal dilation (focal involving | the [0.1] Primary scienosing cholangitis |
| | right hepatic lobe) | 04 Choledocho(thiasis (galistone in duct) |
| 02) | Intrahepatic dutal dilation (focal involving t | ne [6xi Ductal filling defect(s), other than gallsto |
| | left hepatic lobe) | (01 d) Ductal wall thickening or oedema |
| da) | Intrahepatic ductal dilation (involving both | ight [011] Choledochal cyst |
| | and left hepatic lobes) | [61 2] Ductal mass |
| 04) | Extrahepatic ductal dilation | (01 3) Extrinsic mass compressing bile duct(s) |
| 053 | Diffuse ductal dilation (involving both | [disk] Other, specify: |
| | Intrahepatic and extrahepatic ducts) | |
| H. Porta | l/Hepatio vein abnormalities? ✓ all that a | pply: |
| Hot | None | [H7] Hepatic vein thrombosis - malignant |
| нэј | Portal vein enlargement | [Ho] Involvement of the main portal vein |
| H25 | Hepatic vein enlargement | [H9] Involvement of the right portal vein |
| нај | Nonocciusive portal vein thrombosis | [H1 0] Involvement of the left portal vein |
| H41 | Occlusive portal vein thrombosis - bland | [H11] Budd-Chlari syndrome |
| H51 | Hepatic veln thrombosis - bland | [Hillian] Other, specify: |
| неі | Occlusive portal vein thrombosis - maliona | |




| | Protocol Identifier | | Site Identifier | Subject identifier |
|---|---|---|---|---|
| NV | R IMAGING<br>ESTIGATOR<br>RATIVE/COM | RSPONSORE | D/ViiV SUPPORTED ST | UDIES) (Continued) |
| Providence of the second of th | de a textual desc.<br>il interruptions of<br>ution/butcome, ot<br>lonal pages as ne | ription of the liver im<br>liver therapy includi<br>ther contributing fact<br>reded. | raging including relevant medical his<br>ing dates, treatment required to stab<br>ors, alternative etiologies, and any of<br>CRF for narrative description. If the | ilize the reaction,<br>other relevant information. Use |
| IS ENG | (United States/Unglis | ė | | |
| IVE | R IMAGING | RECORD<br>R SPONSORE | D/ViiV SUPPORTED ST | UDIES) (Continued) |
| IVE<br>INV<br>NVE | ER IMAGING<br>ESTIGATOR'S<br>STIGATOR'S | RECORD<br>R SPONSORE<br>SIGNATURE | D/ViiV SUPPORTED STI | |
| IVE<br>INV<br>IVE | ER IMAGING<br>ESTIGATOR'S<br>STIGATOR'S<br>Investigator is accondically qualified<br>from that I have re | RECORD R SPONSORE SIGNATURE countable for this dat d Sub-investigator. | 9 8 79 0 0 0 0 0 0 0 0 0 0 0 0 0 0 0 0 0 0 | or may delegate signature auth |
| IVE<br>INV<br>NVE<br>The it<br>to a n | ER IMAGING<br>ESTIGATOR'S<br>STIGATOR'S<br>Investigator is accondically qualified<br>from that I have re-<br>agues is, to the be- | RECORD R SPONSORE SIGNATURE countable for this dat d Sub-investigator. | ta. However, the Principal Investigat<br>his report for this subject. All informs<br>t, complete and accurate, as of the | or may delegate signature authors as a second or may delegate signature authors as a second or my date below. |

No. of Persons